CLINICAL TRIAL: NCT00932893
Title: Phase 3, Randomized, Open-label Study Of The Efficacy And Safety Of Pf-02341066 Versus Standard Of Care Chemotherapy (Pemetrexed Or Docetaxel) In Patients With Advanced Non-small Cell Lung Cancer (Nsclc) Harboring A Translocation Or Inversion Event Involving The Anaplastic Lymphoma Kinase (Alk) Gene Locus
Brief Title: An Investigational Drug, PF-02341066 Is Being Studied Versus Standard Of Care In Patients With Advanced Non-Small Cell Lung Cancer With A Specific Gene Profile Involving The Anaplastic Lymphoma Kinase (ALK) Gene
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8081007; 2009-012595-27 (EudraCT Number)
Record Dates: First submitted 2009-06-30; First posted 2009-07-03 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung Neoplasms ALK gene crizotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib; Pemetrexed; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-02341066 (Experimental)
  Interventions: Drug: PF-02341066
- Pemetrexed or Docetaxel (Active Comparator): Investigator selection of either pemetrexed or docetaxel as the active comparator
  Interventions: Drug: Pemetrexed; Drug: Docetaxel

INTERVENTIONS:
Drug: PF-02341066 — PF-02341066, 250 mg BID will be administered orally on a continuous schedule
  Arms: PF-02341066
Drug: Pemetrexed — Pemetrexed, 500 mg/m^2, will be administered by i.v. infusion over 10 minutes on Day 1 of each 21-day cycle
  Arms: Pemetrexed or Docetaxel
Drug: Docetaxel — Docetaxel, 75 mg/m^2, will be administered by i.v. infusion over 1 hour on Day 1 of each 21-day cycle
  Arms: Pemetrexed or Docetaxel

SUMMARY:
This is a Phase 3 trial comparing the safety and anti-tumor activity of PF-02341066 versus pemetrexed or docetaxel in patients with advanced non-small cell lung cancer with specific gene profile involving the ALK gene after failure of one previous chemotherapy regimen that included one platinum drug.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven diagnosis of non-small cell lung cancer
* positive for the ALK fusion gene (test provided by a central laboratory)
* must have had disease progression after only one prior chemotherapy and that regimen but must have included one platinum drug
* tumors must be measurable

Exclusion Criteria:

* prior treatment with PF-02341066
* current treatment in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (259):
- United States (115):
  - University of Arkansas for Medical Research, Winthrop Rockefeller Cancer Institute, Little Rock, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - UCSD Medical Center -La Jolla, La Jolla, California
  - Moores UC San Diego Cancer Center, La Jolla, California
  - Drug Shipping Address: [IRB# 10-001530] Ronald Reagan UCLA, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology Oncology, Los Angeles, California
  - UCLA Ophthalmic Oncology Center, Los Angeles, California
  - University of California-Los Angeles, Los Angeles, California
  - Ship Drug To : Kevin Kong- University of California, Irvine-Pharmacy, Orange, California
  - University of California, Irvine-Medical Center, Orange, California
  - Stanford University-Cancer Center, Palo Alto, California
  - UC Davis Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSD Medical Center- Hillcrest, San Diego, California
  - Santa Monica-UCLA Medical Center and Orthopaedic Hospital, Santa Monica, California
  - University of California, Los Angeles, Santa Monica, California
  - Redwood Regional Medical Group, Inc., Santa Rosa, California
  - Drug Shipment: University of Colorado Cancer Center, Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Denver (CTRC), Aurora, Colorado
  - Unviersity of Colorado Hospital, Anschutz Cancer Pavilion, Aurora, Colorado
  - Unviersity of Colorado Hospital, Anschutz Inpatient Pavilion, Aurora, Colorado
  - Kaiser Permanente, Denver, Colorado
  - Kaiser Permanente, Lafayette, Colorado
  - Drug Shipping for Yale; C/O Thomas Ferencz, RPh, BCOP, New Haven, Connecticut
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Clinical Trial Office, New Haven, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Memorial Cancer Institute, Hollywood, Florida
  - Cancer Center of South Florida Foundation, Inc., Lake Worth, Florida
  - Memorial Cancer Institute (West), Pembroke Pines, Florida
  - H Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institution, Atlanta, Georgia
  - Georgia Cancer Specialists-Administrative Annex, Atlanta, Georgia
  - Georgia Cancer Specialists - Stemmer, Decatur, Georgia
  - Georgia Cancer Specialists-Macon, Macon, Georgia
  - Georgia Cancer Specialists-Kennestone, Marietta, Georgia
  - Georgia Cancer Specialists, Sandy Springs, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Hawaii Medical Center East, Honolulu, Hawaii
  - OnCare Hawaii, Inc., Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Ingalls Memorial Hospital (Drug Shipment Only), Harvey, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Monroe Medical Associates, Harvey, Illinois
  - Monroe Medical Associates, Tinley Park, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Ship Drug to: Investigational Drug Services, Indianapolis, Indiana
  - Wishard Memorial Hospital, Indianapolis, Indiana
  - Springmill Medical Clinic, Indianapolis, Indiana
  - Monroe Medical Associates, Munster, Indiana
  - The Community Hospital, Munster, Indiana
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusette General Hospital, Boston, Massachusetts
  - Massachussetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - DFCI/Pharmacy (Drug Shipment Only), Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Lawrence and Idell Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Siteman Cancer Center, City of Saint Peters, Missouri
  - Siteman Cancer Center- West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University, School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - NSLIJ Health System/Monter Cancer Center, Lake Success, New York
  - Memorial Sloan-Kettering Cancer Center: Rockefeller Outpatient Pavilion, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Department of Medicine MSG at SUNY HSC at Syracuse, INC., d/b/a University Physicians, Oneida, New York
  - Department of Medicine MSG at SUNY HSC at Syracuse, INC., d/b/a University Physicians, Oswego, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Department of Medicine MSG at SUNY HSC at Syracuse, INC., d/b/a University Physicians, Syracuse, New York
  - Investigational Drug Service, Pharmacy Department, UNC Hospitals, Chapel Hill, North Carolina
  - UNC Health Care, NC Cancer Hospital Infusion/lnpatient Pharmacy (CHIP), Chapel Hill, North Carolina
  - UNC Hospitals, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Hospital East, Columbus, Ohio
  - The Ohio State University James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - James Care in Kenny, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania at Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center-Shadyside, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vincent Armenio, MD, East Providence, Rhode Island
  - Pharma Resource, East Providence, Rhode Island
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Vanderbilt Cancer Clinic, Nashville, Tennessee
  - The Vanderbilt Chemo Pharmacy, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - The University of Texas, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Investigational Drug Service, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Australia (4):
  - Sydney Cancer Centre, Camperdown, New South Wales
  - Royal Adelaide Hospital, Department of Medical Oncology, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, Division of Haematology and Medical Oncology, East Melbourne, Victoria
  - Department of Medical Oncology, Nedlands, Western Australia
- Brazil (9):
  - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro, Rio de Janeiro
  - Associacao Hospital de Caridade de Ijui, Ijuí, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII Hospital de Cancer de Barretos, Barretos, São Paulo
  - Fundacao Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto do Câncer de São Paulo "Octavio Frias de Oliveira" - ICESP, São Paulo, São Paulo
  - Fundacao Antonio Prudente, São Paulo, São Paulo
- Bulgaria (5):
  - UMBAL "Tsaritsa Yoanna - ISUL", Klinika po onkoterapiya, Sofia, Bulgaria
  - Spetsializirana Bolnitsa za Aktivno Lechenie po Onkologiya, Klinika po himioterapiya, Sofia, Bulgaria
  - MDOZS Plovdiv EOOD; Parvo vatreshno himioterapevtichno otdelenie, Plovdiv
  - MBAL Voennomeditsinska Academia, MMA HAT Sofia, Sofia
  - MDOZS "Dr. Marko Markov", Otdelenie po onkoterapiya i paliativni grizhi, Varna
- Canada (14):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Alberta Health Services, Holy Cross Site, Calgary, Alberta
  - Office of Dr. John McWhae, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Dr. Georges-L. Dumont Regional Hospital, Moncton, New Brunswick
  - Dr. Leon Richard Oncology Centre, Moncton, New Brunswick
  - RSM Durham Regional Cancer Centre, Oshawa, Ontario
  - Dr. Dana Blakolmer and Associates, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Hopital Notre-Dame du Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
- China (9):
  - SUN Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Nanjing Bayi Hospital, Nanjing, Jiangsu
  - Cancer Institute and Hospital Chinese Academy of Medical Sciences and PUMC, Beijing
  - 307 Hospital of PLA, Beijing
  - Shanghai Chest Hospital/Department of Pulmonary Medicine, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Zhongshan Hospital Fudan University / Respiratory Department, Shanghai
  - Shanghai Pulmonary Hospital/Dept. of Oncology, Shanghai
- France (9):
  - Centre Francois Baclesse, Caen
  - Centre Georges-François Leclerc, Dijon
  - Hopital Albert Michallon, Grenoble
  - Pr Fabrice BARLESI, Marseille
  - Centre Antoine Lacassagne, Nice
  - Groupe Hospitalier Cochin, Paris
  - Hopital Tenon / Service de Pneumologie, Paris
  - Centre Rene Gauducheau / Service d'Oncologie Medicale, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Germany (9):
  - Klinikum der Universitaet zu Koeln, Klinik I fuer Innere Medizin, Cologne
  - Universitaetsklinik Carl-Gustav-Carus Dresden, Dresden
  - Westdeutsches Tumorzentrum, Universitaetsklinikum Essen, Innere Klinik - Tumorforschung, Essen
  - Krankenhaus Grosshansdorf, Zentrum fuer Pneumologie und Thoraxchirurgie, Großhansdorf
  - MVZ Prof. Mathey, Pfrof. Schofer GmbH, Hamburg
  - Thoraxklinik am Universitaetsklinikum Heidelberg, Internistische Onkologie der Thoraxtumoren, Heidelberg
  - Klinikum der Universitaet Muenchen, Medizinische Klink - Innenstadt, Pneumologie, München
  - Pius-Hospital Oldenburg, Oldenburg
  - HSK Dr.- Horst-Schmidt-Kliniken, Innere Medizin III Haematologie, Onkologie, Palliativmedizin, Wiesbaden
- Greece (3):
  - University General Hospital of Heraklion/ Department of Clinical Oncology, Heraklion, Crete
  - General Hospital of Thessaloniki Georgios Papanikolaou, Lung Cancer Neoplasia Research Department, Eksochi, Thessaloniki
  - General Hospital of Chest Diseases of Athens "Sotiria", Athens
- Hong Kong (3):
  - Tuen Mun Hospital, Department of Clinical Oncology, Tuenmen, New Territories
  - Division of Respiratory and Critical Care Medicine, Department of Medicine, Queen Mary Hospital, Pokfulam
  - Department of Clinical Oncology, Prince of Wales Hospital, Shatin, New Territories
- Hungary (6):
  - Orszagos Koranyi TBC és Pulmonologiai Intezet, VI. Bronchologia, Budapest
  - Semmelweis Egyetem Pulmonologia Intezet, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum, Tudogyogyaszati Klinika, Debrecen
  - Veszprem Megyei Onkormanyzat Tudogyogyintezete, Farkasgyepű
  - Fejer Megyei Szent Gyorgy Korhaz, Pulmonologiai Osztaly, Székesfehérvár
  - Pest Megyei Tudogyogyintezet, III. Osztaly, Törökbálint
- Ireland (5):
  - Aseptic Compounding Unit, Dublin
  - Department of Medical Oncology, Dublin
  - Department of Medical Oncology, Galway
  - Merlin Park Imaging Centre, Galway
  - Pharmacy Aseptic Service Unit, Galway
- Italy (13):
  - A.O. di Rilievo Nazionale e di Alta Specialita - S. G. Moscati, Avellino
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Oncologia Medica A, Genova
  - Ospedale Versilia, Oncologia Medica, Lido Di Camaiore (LU)
  - Ospedale San Luca, Lucca
  - Dipartimento Oncologia Medica, UO Medicina 1Q A, Unita' Nuovi Farmaci e Terapie Innovative, Milan
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Ospedale Niguarda Ca' Granda Dipartimento Oncologico, SC Divisione di Oncologia Medica Falk, Milan
  - Nuovo Ospedale San Gerardo, Monza
  - Azienda Ospedaliera Universitaria San Luigi Gonzaga, Orbassano (TO)
  - SC Oncologia Medica, Ospedale Santa Maria della Misericordia, Azienda Ospedaliera di Perugia, Perugia
  - Unita' Operativa Complessa di Pneumologia Oncologica I, Padiglione Flaiani, Roma
  - Centro C.O.E.S., A.O. San Giovanni Battista Le Molinette, Torino
- Japan (10):
  - Aichi cancer center central hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Kyushu Cancer Center, Fukuoka, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Okayama University Hospital, Okayama, Okayama-ken
  - Kinki University Hospital, Osakasayama-shi, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Poland (11):
  - Pracownia Optyczna Bozena Lawrynowicz Optyk Dyplomowany, Olsztyn, NAP
  - Centrum Medyczne Ars Medica, Olsztyn, NAP
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn, NAP
  - Pracownia Tomografii Komputerowej "ALL MEDI" Sp. z o.o., Otwock, Poland
  - Klinika Onkologii i Radioterapii, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc, Olsztyn
  - Centralna Izba Przyjec Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - Oddzial Onkologii Klinicznej z Pododdzialem Dziennej Chemioterapii, Poznan
  - Zaklad Diagnostyki Obrazowej, Poznan
  - Lux Med. Sp.z o.o, Warsaw
- Russia (6):
  - Republican Clinical Oncology Dispensary of the Ministry of Health of Tatarstan Republic, Kazan'
  - State Institution "National Cancer Research Center named after N.N. Blokhin' RAMS", Moscow
  - City Clinical Oncology Dispensary, Saint Petersburg
  - Saint-Petersburg State Medical University named after I.P.Pavlov of Roszdrav, Saint Petersburg
  - Research Institute of Pulmonology, Saint-Peterburg
  - State Medical Institution "Oncology Center #2" of Healthcare Department of Krasnodar Region, Sochi
- South Korea (3):
  - National Cancer Center, Center for Lung Cancer, Goyang-si, Gyeonggi-do
  - Seoul National University Hospital / Department of Internal Medicine, Seoul
  - Samsung MedicaCenter,SungkyunkwanUnivSchoolofMedicine,Div. of Hematology-Oncology, Dep. of Medicine, Seoul
- Spain (11):
  - Complexo Hospitalario Universitario A Coruña. Hospital Teresa Herrera (Materno-Infantil), A Coruña, A Coruña
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Del Mar, Barcelona, Barcelona
  - Hospital General Universitari Vall D´Hebron, Barcelona, Barcelona
  - Institut Catala Doncologia - Hospital Duran I Reynals, L'Hospitalet de Llobregat, Barcelona
  - Consorcio Hospitalario Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen Del Rocio, Seville, Sevilla
- Karolinska Universitetssjukhuset, Onkologiska kliniken, Stockholm, Sweden
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Department of Internal Medicine, Taipei
  - Taipei Veterans General Hospital, Chest Department, Taipei
- United Kingdom (9):
  - Royal Marsden Hospital, Sutton, Surrey
  - The Alexandra Hospital, Cheshire
  - Nuffield Health Wessex Hospital, Eastleigh
  - Royal Free Hospital, London
  - Kings College London at Guy's Hospital, London
  - Royal Marsden Hospital, London
  - Christie Hospital NHS Trust, Department of Medical Oncology, Manchester
  - Cancer and Haematology Centre,, Oxford
  - Southampton University Hospitals NHS Trust, Southampton

REFERENCES:
- [Derived] Camidge DR, Kim EE, Usari T, Polli A, Lewis I, Wilner KD. Renal Effects of Crizotinib in Patients With ALK-Positive Advanced NSCLC. J Thorac Oncol. 2019 Jun;14(6):1077-1085. doi: 10.1016/j.jtho.2019.02.015. Epub 2019 Feb 26. PMID 30822515
- [Derived] Wilner KD, Usari T, Polli A, Kim EE. Comparison of cardiovascular effects of crizotinib and chemotherapy in ALK-positive advanced non-small-cell lung cancer. Future Oncol. 2019 Apr;15(10):1097-1103. doi: 10.2217/fon-2018-0869. Epub 2019 Jan 17. PMID 30652510
- [Derived] Yoneda KY, Scranton JR, Cadogan MA, Tassell V, Nadanaciva S, Wilner KD, Stollenwerk NS. Interstitial Lung Disease Associated With Crizotinib in Patients With Advanced Non-Small Cell Lung Cancer: Independent Review of Four PROFILE Trials. Clin Lung Cancer. 2017 Sep;18(5):472-479. doi: 10.1016/j.cllc.2017.03.004. Epub 2017 Mar 14. PMID 28373069
- [Derived] Lin YT, Yu CJ, Yang JC, Shih JY. Anaplastic Lymphoma Kinase (ALK) Kinase Domain Mutation Following ALK Inhibitor(s) Failure in Advanced ALK Positive Non-Small-Cell Lung Cancer: Analysis and Literature Review. Clin Lung Cancer. 2016 Sep;17(5):e77-e94. doi: 10.1016/j.cllc.2016.03.005. Epub 2016 Mar 30. PMID 27130468
- [Derived] Costa DB, Shaw AT, Ou SH, Solomon BJ, Riely GJ, Ahn MJ, Zhou C, Shreeve SM, Selaru P, Polli A, Schnell P, Wilner KD, Wiltshire R, Camidge DR, Crino L. Clinical Experience With Crizotinib in Patients With Advanced ALK-Rearranged Non-Small-Cell Lung Cancer and Brain Metastases. J Clin Oncol. 2015 Jun 10;33(17):1881-8. doi: 10.1200/JCO.2014.59.0539. Epub 2015 Jan 26. PMID 25624436
- [Derived] Lin YT, Wang YF, Yang JC, Yu CJ, Wu SG, Shih JY, Yang PC. Development of renal cysts after crizotinib treatment in advanced ALK-positive non-small-cell lung cancer. J Thorac Oncol. 2014 Nov;9(11):1720-5. doi: 10.1097/JTO.0000000000000326. PMID 25436806
- [Derived] Shaw AT, Kim DW, Nakagawa K, Seto T, Crino L, Ahn MJ, De Pas T, Besse B, Solomon BJ, Blackhall F, Wu YL, Thomas M, O'Byrne KJ, Moro-Sibilot D, Camidge DR, Mok T, Hirsh V, Riely GJ, Iyer S, Tassell V, Polli A, Wilner KD, Janne PA. Crizotinib versus chemotherapy in advanced ALK-positive lung cancer. N Engl J Med. 2013 Jun 20;368(25):2385-94. doi: 10.1056/NEJMoa1214886. Epub 2013 Jun 1. PMID 23724913
- [Derived] Tamiya A, Okamoto I, Miyazaki M, Shimizu S, Kitaichi M, Nakagawa K. Severe acute interstitial lung disease after crizotinib therapy in a patient with EML4-ALK-positive non-small-cell lung cancer. J Clin Oncol. 2013 Jan 1;31(1):e15-7. doi: 10.1200/JCO.2012.43.3730. Epub 2012 Nov 19. No abstract available. PMID 23169500
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081007&StudyName=An%20Investigational%20Drug%2C%20PF-02341066%20Is%20Being%20Studied%20Versus%20Standard%20Of%20Care%20In%20Patients%20With%20Advanced%20Non-Small%20Cell%20Lung%20Cancer%20Wit

RESULTS

PARTICIPANT FLOW:
Groups:
- Crizotinib: Crizotinib (PF-02341066) 250 mg (administered as two 100-mg tablets and one 50-mg tablet) orally twice daily continuously in 21-day cycles. Treatment was continued until disease progression, unacceptable toxicity or withdrawal of consent occurred.
- Chemotherapy: Pemetrexed 500 mg per square meter (mg/m^2) intravenous infusion over 10 minutes or docetaxel 75 mg/m^2 intravenous infusion over 1 hour on Day 1 of 21-day cycle, as per investigator discretion. Treatment was continued until disease progression, unacceptable toxicity or withdrawal of consent occurred.
Period: Overall Study
Arm/Group | Crizotinib | Chemotherapy
Started | 173 | 174
Treated | 172 | 171
Completed | 40 | 4
Not Completed | 133 | 170
Not completed — Death | 115 | 24
Not completed — Lost to Follow-up | 8 | 0
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Other | 5 | 144

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized to study treatment.
Groups:
- Chemotherapy: Pemetrexed 500 mg/m^2 intravenous infusion over 10 minutes or docetaxel 75 mg/m^2 intravenous infusion over 1 hour on Day 1 of 21-day cycle, as per investigator discretion. Treatment was continued until disease progression, unacceptable toxicity or withdrawal of consent occurred.
- Total: Total of all reporting groups
Arm/Group | Crizotinib | Chemotherapy | Total
Number analyzed (Participants) | 173 | 174 | 347
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (13.1) | 49.8 (13.0) | 50.0 (13.0)
Gender [Count of Participants; unit: Participants]
  Female | 98 | 95 | 193
  Male | 75 | 79 | 154

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS: Time in months from randomization to first documentation of objective disease progression as determined by independent radiology review or to death due to any cause, whichever occurred first. PFS was calculated as (first event date minus the date of randomization plus 1) divided by 30.4. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria version 1.1 (RECIST v1.1), as at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: Randomization until progressive disease (PD) or initiation of antitumor therapy in the absence of PD or death, assessed every 6 weeks (up to 112 weeks)
Population: Full analysis set (FAS) included all participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 173 | 174
months | 7.7 [6.0 to 8.8] | 3.0 [2.6 to 4.3]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; P-value was obtained from 1-sided log-rank test stratified by Eastern Cooperative Oncology Group performance status (ECOG PS) score, brain metastases, and prior epidermal growth factor receptor tyrosine kinase inhibitor (EGFR TKI) treatment. The hazard ratio and corresponding 95% confidence interval (CI) from the stratified Cox Proportional Hazards model were also presented; Test type: Superiority or Other; p < 0.0001, Log Rank — To control family-wise Type 1 error, a step-down procedure was applied in following order: PFS, objective response rate (ORR), overall survival (OS), and disease control rate (DCR). Statistical significance: 1-sided at alpha=0.025; Hazard Ratio (HR) = 0.487, 95% CI [0.371 to 0.638]

2. Secondary Outcome: Overall Survival (OS)
Description: OS: Time in months from randomization to date of death due to any cause. OS was calculated as (the death date minus the date of randomization plus 1) divided by 30.4.
Time Frame: Randomization until death (up to 4.5 years)
Population: FAS included all participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 173 | 174
months | 21.7 [18.9 to 30.5] | 21.9 [16.8 to 26.0]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; P-value was obtained from 1-sided log-rank test stratified by ECOG PS score, brain metastases, and prior EGFR TKI treatment. The hazard ratio and corresponding 95% CI from the stratified Cox proportional hazards model were also presented; Test type: Superiority or Other; p = 0.1145, Log Rank — Statistical significance: 1-sided at alpha=0.025; Hazard Ratio (HR) = 0.854, 95% CI [0.661 to 1.104]

3. Secondary Outcome: Overall Survival Probability at Months 6 and 12
Description: Overall survival probability at Month 6 and 12 was defined as the probability of survival at 6 and 12 months respectively, after the randomization of study treatment. The survival probability was estimated using the Kaplan-Meier method.
Time Frame: Month 6, 12
Population: FAS included all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percent chance of survival
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 173 | 174
percent chance of survival
  Month 6 | 86.6 [80.5 to 90.9] | 83.8 [77.4 to 88.5]
  Month 12 | 70.4 [62.9 to 76.7] | 66.7 [59.1 to 73.2]

4. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with objective response based on assessment of complete response (CR) or partial response (PR) according to RECIST v1.1. CR: disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 millimeter [mm] short axis). PR: at least 30 percent (%) decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. Objective response is based on independent radiology review.
Time Frame: Randomization until PD or initiation of antitumor therapy in the absence of PD or death, assessed every 6 weeks (up to 112 weeks)
Population: FAS included all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 173 | 174
percentage of participants | 65.3 [57.7 to 72.4] | 19.5 [13.9 to 26.2]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; P-value was obtained from Cochran-Mantel-Haenszel (CMH) test stratified by ECOG PS, brain metastases, and prior EGFR TKI treatment. The risk ratio and corresponding 95% CI from the stratified CMH test were also reported; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Statistical significance: 2-sided at alpha=0.025; Risk Ratio (RR) = 3.394, 95% CI [2.463 to 4.676]

5. Secondary Outcome: Percentage of Participants With Disease Control at Week 6
Description: Disease control: participants with CR, PR, or stable disease (SD) according to RECIST v1.1. CR: disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 mm short axis). PR: at least 30 % decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. PD: at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. Disease control is based on independent radiology review.
Time Frame: Week 6
Population: FAS included all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 173 | 174
percentage of participants | 81.5 [74.9 to 87.0] | 55.2 [47.5 to 62.7]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; P-value was obtained from CMH test stratified by ECOG PS, brain metastases, and prior EGFR TKI treatment. The risk ratio and corresponding 95% CI from the stratified CMH test were also reported; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Statistical significance: 2-sided at alpha=0.0004; Risk Ratio (RR) = 1.502, 95% CI [1.297 to 1.741]

6. Secondary Outcome: Percentage of Participants With Disease Control at Week 12
Description: Disease control: participants with CR, PR, or SD according to RECIST v1.1. CR: disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 mm short axis). PR: at least 30 % decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: Week 12
Population: FAS included all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 173 | 174
percentage of participants | 64.2 [56.5 to 71.3] | 38.5 [31.2 to 46.2]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Statistical significance: 2-sided at alpha=0.0004; Risk Ratio (RR) = 1.697, 95% CI 2-sided [1.368 to 2.103]

7. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to any cause minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 7.02. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 4
Population: FAS included all participants who were randomized to study treatment. Here 'N' (number of participant analyzed) signifies participants with objective tumor response.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 113 | 34
weeks | 32.1 [26.4 to 42.3] | 24.4 [15 to 36]

8. Secondary Outcome: Time to Tumor Response (TTR)
Description: Time from date of randomization to first documentation of objective tumor response. TTR was calculated for the subgroup of participants with objective tumor response. Objective tumor response was defined as CR or PR according to RECIST v1.1. CR: disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 mm short axis). PR: at least 30 % decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.
Time Frame: as for outcome 4
Population: as for outcome 7
Measure: Median (Full Range); unit: weeks
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 113 | 34
weeks | 6.3 [4.4 to 48.4] | 12.6 [5 to 37.1]

9. Secondary Outcome: Plasma Concentration of Crizotinib
Description: Only participants receiving crizotinib were to be analyzed for this outcome measure as per planned analysis.
Time Frame: Pre-dose on Cycle 1 Day 1, Cycle 1 Day 15, and Day 1 of Cycles 2, 3, 5
Population: Pharmacokinetic (PK) analysis population included all randomized participants who received at least 1 dose of study treatment and had 1 of the PK parameters of interest. Here "N" (number of participants analyzed) signifies participants evaluable for this measure. n=participants evaluable at specific time points.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Crizotinib
Number analyzed (Participants) | 152
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 (n=15) | NA (NA) — Data was not summarized since none of the participants had Ctrough values above lower limit of quantification (LLOQ).
  Cycle 1 Day 15 (n=92) | 298 (148)
  Cycle 2 Day 1 (n=62) | 293 (154)
  Cycle 3 Day 1 (n=61) | 306 (135)
  Cycle 5 Day 1 (n=47) | 291 (156)

10. Secondary Outcome: Number of Participants With Categorical Maximum QTcF for Crizotinib
Description: QT interval corrected using Fridericia's formula (QTcF): QT interval (time corresponding to the beginning of depolarization to re-polarization of the ventricles) divided by cube root of RR interval. Maximum QTcF was categorized as less than (<) 450 milliseconds (msec), 450 msec to <480 msec, 480 msec to <500 msec, and more than or equal to (>=) 500 msec. A participant is reported only once under the maximum QTcF interval observed at any of the time-points. Only participants receiving crizotinib were to be analyzed for this outcome measure as per planned analysis.
Time Frame: Pre-dose on Day 1 of Cycle 1, 2 to 6 hours post-dose on Day 1 of Cycle 1, 2
Population: ECG-evaluable population included all randomized participants who received at least 1 dose of study treatment, and had a baseline and at least 1 post-baseline ECG measurement.
Measure: Number; unit: participants
Arm/Group | Crizotinib
Number analyzed (Participants) | 155
participants
  <450 msec | 137
  450 msec to <480 msec | 9
  480 msec to <500 msec | 1
  >=500 msec | 8

11. Secondary Outcome: Plasma Concentration of Soluble c-Met Ectodomain and Hepatocyte Growth Factor Scatter Proteins
Description: Descriptive statistics (absolute value and change from baseline as measured by ratio to baseline) for each best overall response category (CR, PR, SD, PD or combined) have been used to summarize the data from optional soluble c-Met ectodomain assays for crizotinib treated patients.
Time Frame: Pre-dose on Day 1 of Cycle 1, 2 to 6 hours post-dose on Day 1 of Cycle 2, end of treatment (up to 112 weeks)
Population: The soluble biomarker-evaluable population includes patients from the SA population that received PF-02341066, who have an optional blood sample prior to dosing on Cycle 1 Day 1 and have at least 1 on-treatment soluble biomarker evaluation (Cycle 2 Day 1 and/or end of treatment).
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Overall Values: Overall assessment for complete response, partial response, stable disease, progressive disease and early death
Arm/Group | Overall Values
Number analyzed (Participants) | 172
nanogram per milliliter (ng/mL)
  Baseline (N = 81) | 1428.3 (363.9)
  Cycle 2 Day 1 6-hour post dose (N = 69) | 1683.0 (325.6)
  End of treatment (N = 40) | 1751.8 (327.9)

12. Secondary Outcome: Time to Deterioration (TTD) in Participant Reported Pain, Dyspnea, and Cough
Description: TTD in pain (pain in chest from European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Supplement Module for Lung Cancer [EORTC QLQ-LC13]), dyspnea (from EORTC QLQ-LC13), or cough (from EORTC QLQ-LC13) symptoms was defined as the time from randomization to the earliest time the participant's score showed a 10 point or higher increase from baseline in any of the three symptoms from the instrument. The transformed score of pain, dyspnea, and cough symptom scales of EORTC QLQ-LC13 range from 0 to 100, greater scores = higher symptom severity.
Time Frame: Baseline up to end of treatment (up to 112 weeks)
Population: Patient Reported Outcome (PRO) evaluable population included all randomized participants who received at least 1 dose of study treatment, and had a baseline and at least 1 post-baseline PRO assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 162 | 151
months | 4.5 [3.0 to 6.9] | 1.4 [1.0 to 1.6]
Statistical Analysis 1: Comparison: Crizotinib vs Chemotherapy; The p-value was obtained from 2-sided unstratified log-rank test. The hazard ratio and corresponding 95% CI from the Cox Proportional Hazards model were also presented; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.497, 95% CI [0.373 to 0.661]

13. Secondary Outcome: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30: included global health status/quality of life (QoL), functional scales (physical, role, cognitive, emotional, and social), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulties). Most questions used 4- point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores averaged, transformed to 0-100 scale; higher score for Global Qol/functional scales=better level of QoL/functioning or higher score for symptom scale=greater degree of symptoms.
Time Frame: Baseline, Day (D) 1 of each cycle (C) until disease progression, end of treatment (EOT, up to 112 weeks)
Population: FAS included all participants who were randomized to study treatment. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure and "n" signifies participants who were evaluable for specified time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 165 | 163
units on a scale
  Global QoL: Baseline (n=165, 162) | 57.2 (21.5) | 58.1 (22.2)
  Global QoL: C2D1 (n=154, 133) | 64.5 (21.8) | 58.1 (23.1)
  Global QoL: C3D1 (n=154, 106) | 65.2 (22.1) | 59.4 (23.1)
  Global QoL: C4D1 (n=135, 90) | 68.4 (19.6) | 61.1 (20.8)
  Global QoL: C5D1 (n=123, 74) | 68.5 (20.2) | 64.1 (22.7)
  Global QoL: C6D1 (n=120, 70) | 68.3 (19.8) | 67.5 (23.5)
  Global QoL: C7D1 (n=114, 52) | 69.5 (19.3) | 66.5 (23.1)
  Global QoL: C8D1 (n=110, 43) | 68.7 (20.1) | 66.9 (25.3)
  Global QoL: C9D1 (n=101, 37) | 68.7 (21.0) | 66.4 (27.8)
  Global QoL: C10D1 (n=94, 33) | 67.0 (21.6) | 67.4 (26.8)
  Global QoL: C11D1 (n=83, 25) | 69.5 (20.2) | 71.0 (21.8)
  Global QoL: C12D1 (n=76, 23) | 67.9 (22.0) | 65.6 (24.1)
  Global QoL: C13D1 (n=74, 21) | 66.8 (23.6) | 66.7 (23.6)
  Global QoL: C14D1 (n=66, 19) | 71.5 (20.0) | 65.8 (23.4)
  Global QoL: C15D1 (n=62, 16) | 69.0 (22.2) | 66.1 (24.1)
  Global QoL: C16D1 (n=53, 12) | 69.7 (18.1) | 63.2 (25.5)
  Global QoL: C17D1 (n=47, 11) | 67.6 (20.5) | 69.7 (23.4)
  Global QoL: C18D1 (n=44, 11) | 65.7 (19.9) | 70.5 (22.5)
  Global QoL: C19D1 (n=40, 9) | 69.2 (19.2) | 72.2 (20.0)
  Global QoL: C20D1 (n=35, 8) | 64.3 (20.6) | 60.4 (21.2)
  Global QoL: C21D1 (n=30, 8) | 65.0 (18.4) | 63.5 (23.5)
  Global QoL: C22D1 (n=24, 7) | 70.8 (19.3) | 64.3 (24.9)
  Global QoL: C23D1 (n=23, 4) | 67.0 (22.5) | 50.0 (19.2)
  Global QoL: C24D1 (n=20, 3) | 67.1 (18.8) | 55.6 (19.2)
  Global QoL: C25D1 (n=18, 3) | 67.1 (17.7) | 61.1 (19.2)
  Global QoL: C26D1 (n=14, 3) | 60.7 (22.0) | 55.6 (12.7)
  Global QoL: C27D1 (n=14, 2) | 58.9 (20.3) | 41.7 (0.0)
  Global QoL: C28D1 (n=11, 2) | 66.7 (18.3) | 54.2 (17.7)
  Global QoL: C29D1 (n=8, 2) | 59.4 (18.6) | 41.7 (11.8)
  Global QoL: C30D1 (n=8, 1) | 64.6 (19.3) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Global QoL: C31D1 (n=7, 0) | 64.3 (17.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Global QoL: C32D1 (n=6, 0) | 59.7 (17.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Global QoL: C33D1 (n=6, 0) | 66.7 (18.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Global QoL: C34D1 (n=5, 0) | 68.3 (14.9) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Global QoL: C35D1 (n=4, 0) | 60.4 (22.9) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Global QoL: C36D1 (n=1, 0) | 66.7 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Global QoL: C37D1 (n=1, 0) | 66.7 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Physical Functioning: Baseline (n=165, 163) | 76.3 (20.7) | 75.8 (21.9)
  Physical Functioning: C2D1 (n=155, 133) | 79.2 (20.9) | 73.5 (22.3)
  Physical Functioning: C3D1 (n=154, 106) | 82.3 (18.1) | 75.5 (20.2)
  Physical Functioning: C4D1 (n=135, 91) | 83.8 (16.2) | 76.6 (20.2)
  Physical Functioning: C5D1 (n=123, 74) | 84.5 (16.2) | 78.6 (23.0)
  Physical Functioning: C6D1 (n=120, 70) | 86.2 (16.7) | 80.7 (19.7)
  Physical Functioning: C7D1 (n=115, 52) | 86.7 (15.0) | 80.3 (19.7)
  Physical Functioning: C8D1 (n=111, 43) | 86.5 (16.3) | 81.6 (18.5)
  Physical Functioning: C9D1 (n=101, 37) | 87.7 (14.2) | 82.3 (19.1)
  Physical Functioning: C10D1 (n=94, 33) | 87.9 (14.8) | 81.8 (20.7)
  Physical Functioning: C11D1 (n=84, 25) | 87.2 (16.7) | 83.2 (19.0)
  Physical Functioning: C12D1 (n=76, 23) | 88.1 (15.3) | 79.7 (22.8)
  Physical Functioning: C13D1 (n=74, 21) | 89.3 (13.9) | 78.4 (23.6)
  Physical Functioning: C14D1 (n=66, 19) | 89.0 (14.3) | 80.0 (21.4)
  Physical Functioning: C15D1 (n=62, 16) | 87.8 (15.3) | 82.9 (15.4)
  Physical Functioning: C16D1 (n=53, 12) | 89.3 (11.5) | 81.1 (19.5)
  Physical Functioning: C17D1 (n=47, 11) | 86.6 (16.8) | 81.8 (15.8)
  Physical Functioning: C18D1 (n=45, 11) | 88.4 (13.3) | 82.4 (16.1)
  Physical Functioning: C19D1 (n=40, 9) | 88.3 (12.4) | 81.5 (12.8)
  Physical Functioning: C20D1 (n=35, 8) | 87.6 (12.7) | 79.2 (17.3)
  Physical Functioning: C21D1 (n=30, 8) | 88.4 (10.9) | 77.5 (22.5)
  Physical Functioning: C22D1 (n=24, 7) | 90.6 (8.3) | 78.1 (24.3)
  Physical Functioning: C23D1 (n=23, 4) | 88.0 (13.1) | 60.0 (27.2)
  Physical Functioning: C24D1 (n=20, 3) | 85.0 (14.0) | 64.4 (32.9)
  Physical Functioning: C25D1 (n=18, 3) | 87.4 (11.6) | 60.0 (29.1)
  Physical Functioning: C26D1 (n=14, 3) | 80.5 (25.3) | 62.2 (30.8)
  Physical Functioning: C27D1 (n=14, 2) | 78.6 (27.8) | 50.0 (23.6)
  Physical Functioning: C28D1 (n=11, 2) | 81.8 (24.1) | 60.0 (18.9)
  Physical Functioning: C29D1 (n=8, 2) | 85.0 (15.0) | 46.7 (28.3)
  Physical Functioning: C30D1 (n=8, 1) | 82.5 (21.4) | 26.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Physical Functioning: C31D1 (n=7, 0) | 83.8 (17.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Physical Functioning: C32D1 (n=6, 0) | 88.9 (9.1) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Physical Functioning: C33D1 (n=6, 0) | 90.0 (7.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Physical Functioning: C34D1 (n=5, 0) | 85.3 (7.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Physical Functioning: C35D1 (n=4, 0) | 91.7 (3.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Physical Functioning: C36D1 (n=1, 0) | 86.7 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Physical Functioning: C37D1 (n=1, 0) | 86.7 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Role Functioning: Baseline (n=165, 163) | 69.3 (28.7) | 66.6 (30.2)
  Role Functioning: C2D1 (n=155, 133) | 73.8 (28.9) | 64.7 (29.7)
  Role Functioning: C3D1 (n=154, 106) | 74.4 (28.6) | 65.3 (27.7)
  Role Functioning: C4D1 (n=134, 91) | 77.9 (25.7) | 67.2 (27.3)
  Role Functioning: C5D1 (n=123, 74) | 78.2 (24.3) | 69.6 (27.4)
  Role Functioning: C6D1 (n=120, 70) | 80.0 (24.1) | 69.5 (26.2)
  Role Functioning: C7D1 (n=115, 52) | 81.7 (22.6) | 72.1 (25.9)
  Role Functioning: C8D1 (n=111, 43) | 80.4 (23.9) | 75.2 (28.3)
  Role Functioning: C9D1 (n=101, 37) | 80.9 (25.8) | 76.6 (27.6)
  Role Functioning: C10D1 (n=94, 33) | 81.6 (23.1) | 75.3 (28.3)
  Role Functioning: C11D1 (n=84, 25) | 81.3 (23.8) | 75.3 (25.5)
  Role Functioning: C12D1 (n=76, 23) | 81.6 (23.2) | 72.5 (29.6)
  Role Functioning: C13D1 (n=74, 21) | 80.2 (25.5) | 68.3 (32.0)
  Role Functioning: C14D1 (n=66, 19) | 83.8 (21.3) | 68.4 (30.4)
  Role Functioning: C15D1 (n=62, 16) | 80.6 (24.0) | 77.1 (27.8)
  Role Functioning: C16D1 (n=53, 12) | 84.0 (19.0) | 69.4 (34.0)
  Role Functioning: C17D1 (n=47, 11) | 77.7 (25.4) | 71.2 (38.1)
  Role Functioning: C18D1 (n=45, 11) | 80.0 (22.4) | 71.2 (31.7)
  Role Functioning: C19D1 (n=40, 9) | 82.1 (19.4) | 74.1 (29.0)
  Role Functioning: C20D1 (n=35, 8) | 81.9 (17.8) | 70.8 (36.5)
  Role Functioning: C21D1 (n=30, 8) | 80.0 (24.1) | 66.7 (32.1)
  Role Functioning: C22D1 (n=24, 7) | 84.7 (19.0) | 67.9 (33.5)
  Role Functioning: C23D1 (n=23, 4) | 76.8 (26.9) | 37.5 (25.0)
  Role Functioning: C24D1 (n=20, 3) | 80.8 (24.3) | 44.4 (38.5)
  Role Functioning: C25D1 (n=18, 3) | 87.0 (19.4) | 44.4 (25.5)
  Role Functioning: C26D1 (n=14, 3) | 75.0 (29.1) | 33.3 (33.3)
  Role Functioning: C27D1 (n=14, 2) | 69.0 (35.1) | 25.0 (11.8)
  Role Functioning: C28D1 (n=11, 2) | 77.3 (33.6) | 25.0 (35.4)
  Role Functioning: C29D1 (n=8, 2) | 77.1 (34.4) | 25.0 (11.8)
  Role Functioning: C30D1 (n=8, 1) | 77.1 (34.4) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Role Functioning: C31D1 (n=7, 0) | 71.4 (36.9) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Role Functioning: C32D1 (n=6, 0) | 86.1 (12.5) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Role Functioning: C33D1 (n=6, 0) | 88.9 (13.6) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Role Functioning: C34D1 (n=5, 0) | 96.7 (7.5) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Role Functioning: C35D1 (n=4, 0) | 91.7 (16.7) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Role Functioning: C36D1 (n=1, 0) | 100.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Role Functioning: C37D1 (n=1, 0) | 100.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Emotional Functioning: Baseline (n=165, 162) | 74.5 (21.3) | 73.7 (20.7)
  Emotional Functioning: C2D1 (n=155, 133) | 83.1 (18.7) | 77.7 (19.3)
  Emotional Functioning: C3D1 (n=154, 106) | 83.3 (16.7) | 77.9 (21.5)
  Emotional Functioning: C4D1 (n=135, 90) | 84.1 (17.3) | 80.5 (18.9)
  Emotional Functioning: C5D1 (n=123, 74) | 83.0 (19.1) | 79.8 (19.9)
  Emotional Functioning: C6D1 (n=120, 70) | 85.3 (17.8) | 81.2 (19.4)
  Emotional Functioning: C7D1 (n=115, 52) | 86.4 (16.5) | 81.9 (17.6)
  Emotional Functioning: C8D1 (n=111, 43) | 83.9 (19.8) | 81.6 (20.7)
  Emotional Functioning: C9D1 (n=101, 37) | 84.4 (19.0) | 82.4 (19.6)
  Emotional Functioning: C10D1 (n=94, 33) | 87.2 (16.8) | 81.8 (21.2)
  Emotional Functioning: C11D1 (n=84,25) | 86.1 (16.7) | 85.0 (17.8)
  Emotional Functioning: C12D1 (n=76, 23) | 85.3 (18.6) | 84.8 (18.6)
  Emotional Functioning: C13D1 (n=74, 21) | 84.9 (19.0) | 80.6 (19.1)
  Emotional Functioning: C14D1 (n=66, 19) | 84.5 (19.9) | 81.6 (21.1)
  Emotional Functioning: C15D1 (n=62, 16) | 86.3 (18.0) | 82.3 (18.2)
  Emotional Functioning: C16D1 (n=53, 12) | 85.8 (17.6) | 77.8 (27.8)
  Emotional Functioning: C17D1 (n=47, 11) | 85.6 (22.0) | 79.5 (23.4)
  Emotional Functioning: C18D1 (n=44, 11) | 86.4 (17.2) | 75.8 (27.8)
  Emotional Functioning: C19D1 (n=40, 9) | 87.3 (16.0) | 81.5 (20.7)
  Emotional Functioning: C20D1 (n=35, 8) | 83.8 (17.5) | 82.3 (25.0)
  Emotional Functioning: C21D1 (n=30, 8) | 84.5 (17.1) | 80.2 (29.5)
  Emotional Functioning: C22D1 (n=24, 7) | 83.7 (21.6) | 78.6 (24.9)
  Emotional Functioning: C23D1 (n=23, 4) | 84.1 (19.8) | 70.8 (21.0)
  Emotional Functioning: C24D1 (n=20, 3) | 87.9 (16.1) | 66.7 (30.0)
  Emotional Functioning: C25D1 (n=18, 3) | 81.5 (19.5) | 72.2 (24.1)
  Emotional Functioning: C26D1 (n=14, 3) | 73.2 (28.3) | 72.2 (24.1)
  Emotional Functioning: C27D1 (n=14, 2) | 70.8 (27.3) | 58.3 (0.0)
  Emotional Functioning: C28D1 (n=11, 2) | 81.1 (27.2) | 58.3 (0.0)
  Emotional Functioning: C29D1 (n=8, 2) | 86.5 (15.4) | 54.2 (5.9)
  Emotional Functioning: C30D1 (n=8, 1) | 84.4 (25.0) | 58.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Emotional Functioning: C31D1 (n=7, 0) | 76.2 (28.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Emotional Functioning: C32D1 (n=6, 0) | 87.5 (17.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Emotional Functioning: C33D1 (n=6, 0) | 90.3 (13.4) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Emotional Functioning: C34D1 (n=5, 0) | 91.7 (14.4) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Emotional Functioning: C35D1 (n=4, 0) | 83.3 (20.4) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Emotional Functioning: C36D1 (n=1, 0) | 58.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Emotional Functioning: C37D1 (n=1, 0) | 58.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Cognitive Functioning: Baseline (n=165, 162) | 85.6 (18.3) | 83.6 (22.3)
  Cognitive Functioning: C2D1 (n=155, 133) | 85.5 (18.9) | 84.5 (20.6)
  Cognitive Functioning: C3D1 (n=154, 106) | 87.0 (15.7) | 83.8 (20.4)
  Cognitive Functioning: C4D1 (n=135, 90) | 88.1 (15.6) | 82.6 (20.4)
  Cognitive Functioning: C5D1 (n=123, 74) | 88.9 (14.4) | 82.7 (22.0)
  Cognitive Functioning: C6D1 (n=120, 70) | 87.5 (15.3) | 83.8 (19.2)
  Cognitive Functioning: C7D1 (n=115, 52) | 86.7 (15.6) | 85.3 (18.3)
  Cognitive Functioning: C8D1 (n=111, 43) | 87.8 (14.7) | 82.2 (23.4)
  Cognitive Functioning: C9D1 (n=101, 37) | 88.3 (16.6) | 84.7 (21.7)
  Cognitive Functioning: C10D1 (n=94, 33) | 89.2 (16.0) | 80.8 (22.1)
  Cognitive Functioning: C11D1 (n=84, 25) | 87.9 (14.9) | 85.3 (19.4)
  Cognitive Functioning: C12D1 (n=76, 23) | 89.5 (14.4) | 80.4 (22.8)
  Cognitive Functioning: C13D1 (n=74, 21) | 88.5 (15.6) | 79.4 (27.8)
  Cognitive Functioning: C14D1 (n=66, 19) | 88.9 (14.7) | 81.6 (24.1)
  Cognitive Functioning: C15D1 (n=62, 16) | 87.6 (15.4) | 84.4 (18.7)
  Cognitive Functioning: C16D1 (n=53, 12) | 87.4 (14.2) | 72.2 (25.9)
  Cognitive Functioning: C17D1 (n=47, 11) | 85.1 (15.2) | 75.8 (21.6)
  Cognitive Functioning: C18D1 (n=44, 11) | 88.3 (14.6) | 75.8 (25.1)
  Cognitive Functioning: C19D1 (n=40, 9) | 87.5 (14.5) | 70.4 (23.2)
  Cognitive Functioning: C20D1 (n=35, 8) | 85.7 (15.2) | 72.9 (23.5)
  Cognitive Functioning: C21D1 (n=30, 8) | 85.6 (15.0) | 72.9 (23.5)
  Cognitive Functioning: C22D1 (n=24, 7) | 86.1 (15.3) | 69.0 (24.4)
  Cognitive Functioning: C23D1 (n=23, 4) | 85.5 (14.5) | 58.3 (21.5)
  Cognitive Functioning: C24D1 (n=20, 3) | 85.8 (19.7) | 61.1 (34.7)
  Cognitive Functioning: C25D1 (n=18, 3) | 86.1 (15.4) | 55.6 (25.5)
  Cognitive Functioning: C26D1 (n=14, 3) | 81.0 (26.0) | 61.1 (34.7)
  Cognitive Functioning: C27D1 (n=14, 2) | 76.2 (25.9) | 41.7 (11.8)
  Cognitive Functioning: C28D1 (n=11, 2) | 78.8 (21.2) | 41.7 (11.8)
  Cognitive Functioning: C29D1 (n=8, 2) | 87.5 (11.8) | 33.3 (0.0)
  Cognitive Functioning: C30D1 (n=8, 1) | 83.3 (23.6) | 16.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Cognitive Functioning: C31D1 (n=7, 0) | 81.0 (20.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Cognitive Functioning: C32D1 (n=6, 0) | 83.3 (18.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Cognitive Functioning: C33D1 (n=6, 0) | 86.1 (16.4) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Cognitive Functioning: C34D1 (n=5, 0) | 90.0 (9.1) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Cognitive Functioning: C35D1 (n=4, 0) | 95.8 (8.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Cognitive Functioning: C36D1 (n=1, 0) | 100.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Cognitive Functioning: C37D1 (n=1, 0) | 83.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Social Functioning: Baseline (n=165, 162) | 68.0 (27.7) | 67.1 (29.0)
  Social Functioning: C2D1 (n=155, 133) | 75.9 (25.1) | 69.5 (28.1)
  Social Functioning: C3D1 (n=154, 106) | 78.5 (24.0) | 72.5 (26.7)
  Social Functioning: C4D1 (n=135, 90) | 79.4 (23.9) | 71.7 (26.3)
  Social Functioning: C5D1 (n=123, 74) | 79.4 (23.8) | 74.5 (27.1)
  Social Functioning: C6D1 (n=120, 70) | 81.8 (22.1) | 76.4 (27.3)
  Social Functioning: C7D1 (n=115, 52) | 82.3 (21.8) | 77.9 (24.6)
  Social Functioning: C8D1 (n=111, 43) | 82.0 (21.3) | 77.5 (24.4)
  Social Functioning: C9D1 (n=101, 37) | 80.4 (24.7) | 80.2 (21.8)
  Social Functioning: C10D1 (n=94, 33) | 81.9 (25.1) | 76.3 (27.0)
  Social Functioning: C11D1 (n=84, 25) | 81.9 (23.0) | 78.7 (24.8)
  Social Functioning: C12D1 (n=76, 23) | 82.0 (23.5) | 71.0 (31.9)
  Social Functioning: C13D1 (n=74, 21) | 81.8 (24.7) | 71.4 (28.9)
  Social Functioning: C14D1 (n=66, 19) | 81.3 (23.8) | 69.3 (34.8)
  Social Functioning: C15D1 (n=62, 16) | 81.5 (25.6) | 74.0 (28.5)
  Social Functioning: C16D1 (n=53, 12) | 82.7 (21.9) | 65.3 (35.9)
  Social Functioning: C17D1 (n=47, 11) | 81.9 (24.8) | 69.7 (33.2)
  Social Functioning: C18D1 (n=44, 11) | 82.6 (22.7) | 65.2 (35.3)
  Social Functioning: C19D1 (n=40, 9) | 84.6 (22.8) | 64.8 (31.7)
  Social Functioning: C20D1 (n=35, 8) | 82.9 (23.7) | 70.8 (33.0)
  Social Functioning: C21D1 (n=30, 8) | 82.8 (24.2) | 64.6 (36.1)
  Social Functioning: C22D1 (n=24, 7) | 82.6 (23.8) | 65.5 (39.8)
  Social Functioning: C23D1 (n=23, 4) | 84.4 (23.9) | 41.7 (50.0)
  Social Functioning: C24D1 (n=20, 3) | 84.2 (27.3) | 61.1 (53.6)
  Social Functioning: C25D1 (n=18, 3) | 89.8 (19.1) | 50.0 (50.0)
  Social Functioning: C26D1 (n=14, 3) | 78.6 (28.8) | 50.0 (50.0)
  Social Functioning: C27D1 (n=14, 2) | 85.7 (15.8) | 33.3 (47.1)
  Social Functioning: C28D1 (n=11, 2) | 83.3 (26.9) | 33.3 (47.1)
  Social Functioning: C29D1 (n=8, 2) | 83.3 (25.2) | 33.3 (47.1)
  Social Functioning: C30D1 (n=8, 1) | 85.4 (24.3) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Social Functioning: C31D1 (n=7, 0) | 73.8 (38.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Social Functioning: C32D1 (n=6, 0) | 83.3 (18.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Social Functioning: C33D1 (n=6, 0) | 94.4 (13.6) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Social Functioning: C34D1 (n=5, 0) | 96.7 (7.5) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Social Functioning: C35D1 (n=4, 0) | 91.7 (16.7) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Social Functioning: C36D1 (n=1, 0) | 66.7 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Social Functioning: C37D1 (n=1, 0) | 66.7 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Fatigue: Baseline (n=165, 163) | 38.3 (24.4) | 36.1 (25.3)
  Fatigue: C2D1 (n=155, 133) | 31.4 (23.4) | 39.5 (24.8)
  Fatigue: C3D1 (n=154, 106) | 30.8 (24.1) | 39.4 (24.5)
  Fatigue: C4D1 (n=135, 91) | 27.1 (22.3) | 34.1 (22.1)
  Fatigue: C5D1 (n=123, 74) | 24.7 (19.8) | 31.5 (25.2)
  Fatigue: C6D1 (n=120, 70) | 24.6 (19.3) | 31.0 (22.8)
  Fatigue: C7D1 (n=115, 52) | 23.9 (19.8) | 27.6 (23.1)
  Fatigue: C8D1 (n=111, 43) | 23.2 (18.9) | 26.6 (23.6)
  Fatigue: C9D1 (n=101, 37) | 22.9 (21.7) | 28.5 (26.6)
  Fatigue: C10D1 (n=94, 33) | 21.4 (20.0) | 28.6 (27.9)
  Fatigue: C11D1 (n=84, 25) | 22.1 (19.6) | 22.2 (22.9)
  Fatigue: C12D1 (n=76, 23) | 21.9 (22.9) | 26.1 (24.1)
  Fatigue: C13D1 (n=74, 21) | 23.3 (21.3) | 27.5 (25.2)
  Fatigue: C14D1 (n=66, 19) | 21.7 (21.7) | 28.1 (26.8)
  Fatigue: C15D1 (n=62, 16) | 20.8 (22.5) | 24.3 (24.8)
  Fatigue: C16D1 (n=53, 12) | 22.2 (18.0) | 24.1 (21.6)
  Fatigue: C17D1 (n=47, 11) | 23.4 (20.0) | 23.2 (23.0)
  Fatigue: C18D1 (n=45, 11) | 21.5 (18.3) | 27.3 (22.4)
  Fatigue: C19D1 (n=40, 9) | 20.8 (18.7) | 24.7 (20.6)
  Fatigue: C20D1 (n=35, 8) | 24.4 (19.2) | 27.8 (26.6)
  Fatigue: C21D1 (n=30, 8) | 23.9 (17.8) | 25.7 (27.7)
  Fatigue: C22D1 (n=24, 7) | 23.6 (16.2) | 27.0 (23.9)
  Fatigue: C23D1 (n=23, 4) | 25.1 (19.3) | 47.2 (14.0)
  Fatigue: C24D1 (n=20, 3) | 24.4 (18.9) | 40.7 (23.1)
  Fatigue: C25D1 (n=18, 3) | 24.7 (16.0) | 44.4 (19.2)
  Fatigue: C26D1 (n=14, 3) | 30.2 (25.6) | 44.4 (19.2)
  Fatigue: C27D1 (n=14, 2) | 35.7 (25.1) | 55.6 (15.7)
  Fatigue: C28D1 (n=11, 2) | 28.3 (22.4) | 38.9 (7.9)
  Fatigue: C29D1 (n=8, 2) | 30.6 (22.8) | 50.0 (23.6)
  Fatigue: C30D1 (n=8, 1) | 26.4 (24.4) | 55.6 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Fatigue: C31D1 (n=7, 0) | 28.6 (16.8) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Fatigue: C32D1 (n=6, 0) | 25.9 (5.7) | NA (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Fatigue: C33D1 (n=6, 0) | 18.5 (11.5) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Fatigue: C34D1 (n=5, 0) | 15.6 (16.9) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Fatigue: C35D1 (n=4, 0) | 27.8 (14.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Fatigue: C36D1 (n=1, 0) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Fatigue: C37D1 (n=1, 0) | 11.1 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Nausea and Vomiting: Baseline (n=165, 163) | 8.4 (14.4) | 11.7 (18.0)
  Nausea and Vomiting: C2D1 (n=155, 133) | 15.2 (20.9) | 12.7 (19.0)
  Nausea and Vomiting: C3D1 (n=154, 106) | 13.9 (21.2) | 9.9 (16.6)
  Nausea and Vomiting: C4D1 (n=135, 91) | 9.9 (18.1) | 8.1 (14.1)
  Nausea and Vomiting: C5D1 (n=123, 74) | 9.2 (14.7) | 9.0 (16.8)
  Nausea and Vomiting: C6D1 (n=120, 70) | 10.1 (15.2) | 6.9 (13.2)
  Nausea and Vomiting: C7D1 (n=115, 52) | 7.1 (11.9) | 7.7 (11.7)
  Nausea and Vomiting: C8D1 (n=111, 43) | 8.8 (13.7) | 8.9 (14.7)
  Nausea and Vomiting: C9D1 (n=101, 37) | 6.9 (13.0) | 9.5 (19.9)
  Nausea and Vomiting: C10D1 (n=94, 33) | 8.5 (14.6) | 8.1 (15.7)
  Nausea and Vomiting: C11D1 (n=84, 25) | 8.3 (12.8) | 8.0 (16.0)
  Nausea and Vomiting: C12D1 (n=76, 23) | 6.4 (12.8) | 7.2 (15.8)
  Nausea and Vomiting: C13D1 (n=74, 21) | 8.6 (14.1) | 7.1 (16.3)
  Nausea and Vomiting: C14D1 (n=66, 19) | 5.8 (13.9) | 7.0 (14.0)
  Nausea and Vomiting: C15D1 (n=62, 16) | 5.9 (11.3) | 6.2 (13.4)
  Nausea and Vomiting: C16D1 (n=53, 12) | 5.3 (9.7) | 6.9 (11.1)
  Nausea and Vomiting: C17D1 (n=47, 11) | 7.8 (12.5) | 10.6 (11.2)
  Nausea and Vomiting: C18D1 (n=45, 11) | 7.0 (13.5) | 3.0 (6.7)
  Nausea and Vomiting: C19D1 (n=40, 9) | 8.8 (14.6) | 9.3 (12.1)
  Nausea and Vomiting: C20D1 (n=35, 8) | 7.4 (13.5) | 10.4 (15.3)
  Nausea and Vomiting: C21D1 (n=30, 8) | 7.8 (12.9) | 8.3 (12.6)
  Nausea and Vomiting: C22D1 (n=24, 7) | 2.8 (6.3) | 14.3 (17.8)
  Nausea and Vomiting: C23D1 (n=23, 4) | 5.4 (10.5) | 45.8 (21.0)
  Nausea and Vomiting: C24D1 (n=20, 3) | 7.5 (14.8) | 33.3 (28.9)
  Nausea and Vomiting: C25D1 (n=18, 3) | 3.7 (9.1) | 27.8 (25.5)
  Nausea and Vomiting: C26D1 (n=14, 3) | 10.7 (27.4) | 33.3 (16.7)
  Nausea and Vomiting: C27D1 (n=14, 2) | 11.9 (27.3) | 33.3 (23.6)
  Nausea and Vomiting: C28D1 (n=11, 2) | 3.0 (6.7) | 25.0 (11.8)
  Nausea and Vomiting: C29D1 (n=8, 2) | 10.4 (15.3) | 25.0 (11.8)
  Nausea and Vomiting: C30D1 (n=8, 1) | 6.3 (12.4) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Nausea and Vomiting: C31D1 (n=7, 0) | 14.3 (17.8) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Nausea and Vomiting: C32D1 (n=6, 0) | 11.1 (17.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Nausea and Vomiting: C33D1 (n=6, 0) | 11.1 (17.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Nausea and Vomiting: C34D1 (n=5, 0) | 13.3 (18.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Nausea and Vomiting: C35D1 (n=4, 0) | 12.5 (16.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Nausea and Vomiting: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Nausea and Vomiting: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain: Baseline (n=165, 163) | 23.9 (24.7) | 28.0 (27.3)
  Pain: C2D1 (n=155, 133) | 13.9 (19.8) | 25.7 (25.3)
  Pain: C3D1 (n=154, 106) | 13.7 (20.4) | 23.3 (26.6)
  Pain: C4D1 (n=135, 91) | 13.0 (19.5) | 19.0 (21.5)
  Pain: C5D1 (n=123, 74) | 11.5 (16.7) | 20.5 (23.0)
  Pain: C6D1 (n=120, 70) | 10.6 (15.0) | 19.5 (23.0)
  Pain: C7D1 (n=115, 52) | 9.6 (14.3) | 21.5 (24.3)
  Pain: C8D1 (n=111, 43) | 11.3 (18.0) | 17.4 (23.6)
  Pain: C9D1 (n=101, 37) | 11.8 (18.8) | 23.0 (27.6)
  Pain: C10D1 (n=94, 33) | 8.7 (14.0) | 24.2 (28.6)
  Pain: C11D1 (n=84, 25) | 10.5 (16.3) | 22.0 (27.9)
  Pain: C12D1 (n=76, 23) | 8.6 (14.3) | 25.4 (29.7)
  Pain: C13D1 (n=74, 21) | 10.1 (15.3) | 27.8 (30.4)
  Pain: C14D1 (n=66, 19) | 8.1 (12.8) | 23.7 (26.2)
  Pain: C15D1 (n=62, 16) | 9.4 (15.6) | 22.9 (25.7)
  Pain: C16D1 (n=53, 12) | 9.4 (14.4) | 31.9 (28.8)
  Pain: C17D1 (n=47, 11) | 10.6 (16.1) | 24.2 (27.2)
  Pain: C18D1 (n=45, 11) | 11.1 (18.1) | 24.2 (29.2)
  Pain: C19D1 (n=40, 9) | 11.3 (17.0) | 24.1 (20.6)
  Pain: C20D1 (n=35, 8) | 11.9 (18.8) | 22.9 (28.1)
  Pain: C21D1 (n=30, 8) | 11.7 (15.3) | 29.2 (30.5)
  Pain: C22D1 (n=24, 7) | 6.9 (12.9) | 33.3 (28.9)
  Pain: C23D1 (n=23, 4) | 9.1 (16.1) | 33.3 (36.0)
  Pain: C24D1 (n=20, 3) | 4.2 (11.9) | 27.8 (48.1)
  Pain: C25D1 (n=18, 3) | 4.6 (7.7) | 38.9 (41.9)
  Pain: C26D1 (n=14, 3) | 17.9 (27.3) | 38.9 (41.9)
  Pain: C27D1 (n=14, 2) | 13.1 (25.5) | 58.3 (35.4)
  Pain: C28D1 (n=11, 2) | 4.5 (7.8) | 50.0 (47.1)
  Pain: C29D1 (n=8, 2) | 2.1 (5.9) | 41.7 (35.4)
  Pain: C30D1 (n=8, 1) | 4.2 (7.7) | 83.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pain: C31D1 (n=7, 0) | 4.8 (8.1) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain: C32D1 (n=6, 0) | 5.6 (8.6) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain: C33D1 (n=6, 0) | 2.8 (6.8) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain: C34D1 (n=5, 0) | 3.3 (7.5) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain: C35D1 (n=4, 0) | 8.3 (16.7) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dyspnea: Baseline (n=165, 163) | 31.1 (28.3) | 32.5 (28.2)
  Dyspnea: C2D1 (n=155, 133) | 21.5 (21.4) | 33.6 (27.7)
  Dyspnea: C3D1 (n=154, 106) | 21.6 (23.0) | 33.3 (28.4)
  Dyspnea: C4D1 (n=135, 91) | 17.3 (20.7) | 29.3 (26.2)
  Dyspnea: C5D1 (n=123, 74) | 16.0 (20.6) | 29.3 (24.0)
  Dyspnea: C6D1 (n=120, 70) | 15.8 (22.0) | 26.2 (24.7)
  Dyspnea: C7D1 (n=115, 52) | 17.4 (20.9) | 28.2 (22.3)
  Dyspnea: C8D1 (n=111, 43) | 15.8 (19.7) | 22.5 (28.8)
  Dyspnea: C9D1 (n=101, 37) | 13.9 (19.0) | 23.4 (24.7)
  Dyspnea: C10D1 (n=94, 33) | 17.7 (20.6) | 24.2 (22.5)
  Dyspnea: C11D1 (n=84, 25) | 17.5 (22.8) | 25.3 (22.1)
  Dyspnea: C12D1 (n=76, 23) | 14.5 (19.9) | 30.4 (28.3)
  Dyspnea: C13D1 (n=74, 21) | 14.0 (20.6) | 23.8 (23.9)
  Dyspnea: C14D1 (n=66, 19) | 15.2 (21.2) | 29.8 (24.6)
  Dyspnea: C15D1 (n=62, 16) | 15.6 (21.5) | 20.8 (20.6)
  Dyspnea: C16D1 (n=53, 12) | 13.8 (17.8) | 19.4 (22.3)
  Dyspnea: C17D1 (n=46, 11) | 14.5 (20.7) | 24.2 (21.6)
  Dyspnea: C18D1 (n=45, 11) | 14.1 (16.6) | 24.2 (26.2)
  Dyspnea: C19D1 (n=40, 9) | 14.2 (18.3) | 25.9 (22.2)
  Dyspnea: C20D1 (n=35, 8) | 10.5 (17.7) | 33.3 (25.2)
  Dyspnea: C21D1 (n=30, 8) | 13.3 (16.6) | 33.3 (17.8)
  Dyspnea: C22D1 (n=24, 7) | 13.9 (19.5) | 28.6 (23.0)
  Dyspnea: C23D1 (n=23, 4) | 9.4 (14.9) | 41.7 (16.7)
  Dyspnea: C24D1 (n=20, 3) | 18.3 (20.2) | 44.4 (19.2)
  Dyspnea: C25D1 (n=18, 3) | 11.1 (16.2) | 33.3 (33.3)
  Dyspnea: C26D1 (n=14, 3) | 14.3 (28.4) | 33.3 (33.3)
  Dyspnea: C27D1 (n=14, 2) | 11.9 (16.6) | 50.0 (23.6)
  Dyspnea: C28D1 (n=11, 2) | 12.1 (16.8) | 50.0 (23.6)
  Dyspnea: C29D1 (n=8, 2) | 4.2 (11.8) | 50.0 (23.6)
  Dyspnea: C30D1 (n=8, 1) | 8.3 (15.4) | 66.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Dyspnea: C31D1 (n=7, 0) | 9.5 (16.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dyspnea: C32D1 (n=6, 0) | 16.7 (18.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dyspnea: C33D1 (n=6, 0) | 11.1 (17.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dyspnea: C34D1 (n=5, 0) | 13.3 (18.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dyspnea: C35D1 (n=4, 0) | 16.7 (19.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dyspnea: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dyspnea: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Insomnia : Baseline (n=164, 163) | 22.6 (26.4) | 27.8 (27.3)
  Insomnia : C2D1 (n=155, 133) | 15.3 (23.5) | 27.1 (25.3)
  Insomnia : C3D1 (n=154, 106) | 16.2 (26.2) | 23.6 (26.0)
  Insomnia : C4D1 (n=135, 91) | 13.3 (21.2) | 23.8 (26.9)
  Insomnia : C5D1 (n=123, 74) | 13.6 (21.3) | 25.7 (26.8)
  Insomnia : C6D1 (n=120, 70) | 14.2 (21.9) | 23.3 (25.0)
  Insomnia : C7D1 (n=114, 52) | 9.4 (17.5) | 21.8 (25.5)
  Insomnia : C8D1 (n=111, 43) | 12.5 (21.5) | 21.7 (22.9)
  Insomnia : C9D1 (n=100, 37) | 12.3 (21.5) | 22.5 (24.9)
  Insomnia : C10D1 (n=94, 33) | 13.5 (23.6) | 24.2 (25.4)
  Insomnia : C11D1 (n=84, 25) | 13.9 (22.1) | 22.7 (24.9)
  Insomnia : C12D1 (n=76, 23) | 13.6 (21.9) | 23.2 (25.5)
  Insomnia : C13D1 (n=74, 21) | 10.8 (19.2) | 25.4 (25.6)
  Insomnia : C14D1 (n=66, 19) | 11.1 (18.8) | 24.6 (29.1)
  Insomnia : C15D1 (n=62, 16) | 11.3 (20.0) | 29.2 (26.9)
  Insomnia : C16D1 (n=53, 11) | 13.8 (20.1) | 21.2 (22.5)
  Insomnia : C17D1 (n=47, 11) | 13.5 (21.6) | 15.2 (22.9)
  Insomnia : C18D1 (n=45, 11) | 12.6 (17.8) | 21.2 (27.0)
  Insomnia : C19D1 (n=40, 9) | 13.3 (19.7) | 22.2 (28.9)
  Insomnia : C20D1 (n=35, 8) | 15.2 (20.4) | 20.8 (24.8)
  Insomnia : C21D1 (n=30, 8) | 12.2 (18.5) | 29.2 (27.8)
  Insomnia : C22D1 (n=24, 7) | 12.5 (19.2) | 31.0 (24.4)
  Insomnia : C23D1 (n=23, 4) | 17.4 (26.3) | 50.0 (19.2)
  Insomnia : C24D1 (n=20, 3) | 11.7 (22.4) | 22.2 (38.5)
  Insomnia : C25D1 (n=18, 3) | 20.4 (30.5) | 44.4 (19.2)
  Insomnia : C26D1 (n=14, 3) | 21.4 (33.6) | 22.2 (38.5)
  Insomnia : C27D1 (n=14, 2) | 16.7 (21.7) | 50.0 (23.6)
  Insomnia : C28D1 (n=11, 2) | 9.1 (15.6) | 50.0 (23.6)
  Insomnia : C29D1 (n=8, 2) | 8.3 (15.4) | 33.0 (0.0)
  Insomnia : C30D1 (n=8, 1) | 12.5 (24.8) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Insomnia : C31D1 (n=7, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Insomnia : C32D1 (n=6, 0) | 5.6 (13.6) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Insomnia : C33D1 (n=6, 0) | 5.6 (13.6) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Insomnia : C34D1 (n=5, 0) | 13.3 (18.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Insomnia : C35D1 (n=4, 0) | 16.7 (19.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Insomnia : C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Insomnia : C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Appetite loss : Baseline(n=165, 163) | 24.4 (28.8) | 23.3 (28.2)
  Appetite loss : C2/D1(n=155, 133) | 21.1 (30.2) | 24.3 (28.5)
  Appetite loss : C3/D1(n=154, 106) | 18.4 (29.0) | 21.7 (27.2)
  Appetite loss : C4/D1(n=135, 91) | 14.6 (24.3) | 19.4 (23.3)
  Appetite loss : C5/D1(n=123, 74) | 12.7 (22.4) | 19.4 (28.1)
  Appetite loss : C6/D1(n=120, 70) | 13.6 (21.8) | 12.9 (23.6)
  Appetite loss : C7/D1(n=115, 52) | 10.4 (19.4) | 12.8 (22.0)
  Appetite loss : C8/D1(n=111, 43) | 12.8 (20.8) | 10.9 (22.7)
  Appetite loss : C9/D1(n=101, 37) | 12.2 (239) | 14.4 (27.8)
  Appetite loss : C10/D1(n=94, 33) | 12.4 (22.9) | 14.1 (25.0)
  Appetite loss : C11/D1(n=84, 25) | 13.5 (19.4) | 14.7 (25.6)
  Appetite loss : C12/D1(n=76, 23) | 11.0 (21.4) | 14.5 (24.3)
  Appetite loss : C13/D1(n=74, 21) | 9.5 (20.3) | 17.5 (27.1)
  Appetite loss : C15/D1(n=62, 16) | 8.6 (20.9) | 12.5 (26.9)
  Appetite loss : C16/D1(n=53, 12) | 8.8 (18.7) | 16.7 (30.2)
  Appetite loss : C17/D1(n=47, 11) | 8.5 (16.3) | 15.2 (31.1)
  Appetite loss : C18/D1(n=45, 11) | 11.1 (17.4) | 12.1 (22.5)
  Appetite loss : C19/D1(n=40, 9) | 8.3 (16.5) | 18.5 (33.8)
  Appetite loss : C20/D1(n=35, 8) | 7.6 (16.3) | 20.8 (35.4)
  Appetite loss : C21/D1(n=30, 8) | 11.1 (16.0) | 25.0 (34.5)
  Appetite loss : C22/D1(n=24, 7) | 6.9 (13.8) | 14.3 (37.8)
  Appetite loss : C23/D1(n=23, 4) | 9.4 (14.9) | 50.0 (43.0)
  Appetite loss : C24/D1(n=20, 3) | 5.0 (12.2) | 33.3 (33.3)
  Appetite loss : C25/D1(n=18, 3) | 1.9 (7.9) | 44.4 (50.9)
  Appetite loss : C26/D1(n=14, 3) | 11.9 (21.1) | 33.3 (33.3)
  Appetite loss : C27/D1(n=14, 2) | 7.1 (19.3) | 33.3 (47.1)
  Appetite loss : C28/D1(n=11, 2) | 15.2 (17.4) | 33.3 (47.1)
  Appetite loss : C29/D1(n=8, 2) | 12.5 (17.3) | 33.3 (47.1)
  Appetite loss : C30/D1(n=8, 1) | 8.3 (15.4) | 100.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Appetite loss : C31/D1(n=7, 0) | 14.3 (17.8) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Constipation: Baseline (n=164, 162) | 14.8 (25.1) | 16.9 (25.0)
  Constipation: C2D1 (n=155, 133) | 28.6 (30.5) | 14.0 (24.3)
  Constipation: C3D1 (n=154, 106) | 27.1 (30.0) | 16.0 (22.2)
  Constipation: C4D1 (n=134, 90) | 22.9 (26.6) | 14.8 (25.5)
  Constipation: C5D1 (n=123, 74) | 21.4 (25.7) | 20.3 (29.6)
  Constipation: C6D1 (n=120, 70) | 21.7 (23.9) | 15.7 (23.2)
  Constipation: C7D1 (n=115, 52) | 21.7 (26.1) | 19.9 (26.6)
  Constipation: C8D1 (n=111, 43) | 18.6 (24.1) | 16.3 (24.5)
  Constipation: C9D1 (n=101, 37) | 18.8 (22.3) | 16.2 (21.7)
  Constipation: C10D1 (n=94, 33) | 16.0 (22.8) | 19.2 (25.0)
  Constipation: C11D1 (n=84, 25) | 21.0 (25.8) | 21.3 (19.0)
  Constipation: C12D1 (n=76, 23) | 19.7 (24.5) | 21.7 (23.8)
  Constipation: C13D1 (n=74, 21) | 21.2 (26.2) | 22.2 (26.5)
  Constipation: C14D1 (n=66, 19) | 21.7 (27.1) | 24.6 (31.1)
  Constipation: C15D1 (n=62, 16) | 22.6 (27.5) | 18.7 (21.0)
  Constipation: C16D1 (n=53, 12) | 19.5 (26.5) | 22.2 (25.9)
  Constipation: C17D1 (n=47, 11) | 22.0 (27.2) | 24.2 (30.2)
  Constipation: C18D1 (n=44, 11) | 22.7 (25.7) | 15.2 (22.9)
  Constipation: C19D1 (n=40, 9) | 25.0 (25.9) | 22.2 (23.6)
  Constipation: C20D1 (n=35, 8) | 22.9 (26.5) | 20.8 (24.8)
  Constipation: C21D1 (n=30, 8) | 24.4 (28.9) | 16.7 (25.2)
  Constipation: C22D1 (n=24, 7) | 18.1 (24.0) | 19.0 (26.2)
  Constipation: C23D1 (n=23, 4) | 11.6 (19.1) | 25.0 (31.9)
  Constipation: C24D1 (n=20, 3) | 21.7 (24.8) | 22.2 (19.2)
  Constipation: C25D1 (n=18, 3) | 22.2 (32.3) | 33.3 (33.3)
  Constipation: C26D1 (n=14, 3) | 26.2 (32.5) | 44.4 (50.9)
  Constipation: C27D1 (n=14, 2) | 35.7 (40.2) | 50.0 (23.6)
  Constipation: C28D1 (n=11, 2) | 21.2 (16.8) | 50.0 (23.6)
  Constipation: C29D1 (n=8, 2) | 29.2 (21.4) | 50.0 (23.6)
  Constipation: C30D1 (n=8, 1) | 29.2 (27.8) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Constipation: C31D1 (n=7, 0) | 33.3 (27.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Constipation: C32D1 (n=6, 0) | 33.3 (42.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Constipation: C33D1 (n=6, 0) | 38.9 (25.1) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Constipation: C34D1 (n=5, 0) | 40.0 (43.5) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Constipation: C35D1 (n=4, 0) | 33.3 (27.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Constipation: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Constipation: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Constipation: EOT (n=49, 90) | 28.6 (27.2) | 18.1 (25.6)
  Diarrhea: Baseline (n=165, 162) | 9.7 (19.1) | 7.8 (16.0)
  Diarrhea: C2D1 (n=155, 132) | 18.1 (26.7) | 11.1 (20.5)
  Diarrhea: C3D1 (n=153, 106) | 21.6 (28.7) | 7.9 (18.1)
  Diarrhea: C4D1 (n=134, 90) | 23.1 (26.9) | 8.5 (18.4)
  Diarrhea: C5D1 (n=123, 74) | 24.4 (25.6) | 5.9 (15.0)
  Diarrhea: C6D1 (n=120, 70) | 22.2 (26.4) | 7.1 (16.9)
  Diarrhea: C7D1 (n=115, 52) | 20.6 (24.8) | 9.6 (16.6)
  Diarrhea: C8D1 (n=111, 43) | 18.6 (24.1) | 9.3 (19.7)
  Diarrhea: C9D1 (n=101, 37) | 17.3 (22.8) | 7.2 (16.0)
  Diarrhea: C10D1 (n=94, 33) | 17.7 (22.3) | 7.1 (16.2)
  Diarrhea: C11D1 (n=84, 25) | 21.0 (22.4) | 8.0 (17.4)
  Diarrhea: C12D1 (n=76, 23) | 17.5 (25.2) | 8.7 (15.0)
  Diarrhea: C13D1 (n=74, 21) | 17.6 (23.6) | 12.7 (19.7)
  Diarrhea: C14D1 (n=66, 19) | 17.7 (22.8) | 8.8 (18.7)
  Diarrhea: C15D1 (n=62, 16) | 16.1 (21.5) | 4.2 (11.4)
  Diarrhea: C16D1 (n=52, 12) | 16.0 (20.3) | 5.6 (13.0)
  Diarrhea: C17D1 (n=47, 11) | 19.9 (22.7) | 12.1 (22.5)
  Diarrhea: C18D1 (n=44, 11) | 22.7 (25.7) | 12.1 (22.5)
  Diarrhea: C19D1 (n=40, 9) | 21.7 (25.7) | 7.4 (14.7)
  Diarrhea: C20D1 (n=35, 8) | 21.0 (24.4) | 4.2 (11.8)
  Diarrhea: C21D1 (n=30, 8) | 22.2 (22.0) | 8.3 (15.4)
  Diarrhea: C22D1 (n=24, 7) | 23.6 (25.0) | 11.9 (15.9)
  Diarrhea: C23D1 (n=23, 4) | 15.9 (19.8) | 25.0 (16.7)
  Diarrhea: C24D1 (n=20, 3) | 21.7 (22.4) | 11.1 (19.2)
  Diarrhea: C25D1 (n=18, 3) | 20.4 (25.9) | 22.2 (19.2)
  Diarrhea: C26D1 (n=14, 3) | 19.0 (25.2) | 11.1 (19.2)
  Diarrhea: C27D1 (n=14, 2) | 23.8 (30.5) | 16.7 (23.6)
  Diarrhea: C28D1 (n=11, 2) | 15.2 (17.4) | 16.7 (23.6)
  Diarrhea: C29D1 (n=8, 2) | 20.8 (24.8) | 16.7 (23.6)
  Diarrhea: C30D1 (n=8, 1) | 12.5 (17.3) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Diarrhea: C31D1 (n=7, 0) | 14.3 (17.8) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Diarrhea: C32D1 (n=6, 0) | 11.1 (17.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Diarrhea: C33D1 (n=6, 0) | 11.1 (17.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Diarrhea: C34D1 (n=5, 0) | 6.7 (14.9) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Diarrhea: C35D1 (n=4, 0) | 16.7 (19.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Diarrhea: C36D1 (n=1, 0) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Diarrhea: C37D1 (n=1, 0) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Diarrhea: EOT (n=49, 90) | 18.4 (23.6) | 10.0 (21.5)
  Financial Difficulties: Baseline (n=165, 161) | 28.5 (33.0) | 27.3 (30.7)
  Financial Difficulties: C2D1 (n=155, 133) | 21.9 (27.2) | 22.3 (28.9)
  Financial Difficulties: C3D1 (n=154, 105) | 19.0 (26.6) | 20.3 (27.9)
  Financial Difficulties: C4D1 (n=135, 90) | 17.5 (26.0) | 21.9 (26.0)
  Financial Difficulties: C5D1 (n=123, 74) | 16.8 (25.0) | 19.4 (23.4)
  Financial Difficulties: C6D1 (n=120, 70) | 15.6 (24.0) | 18.6 (25.1)
  Financial Difficulties: C7D1 (n=115, 52) | 14.8 (21.3) | 18.6 (25.9)
  Financial Difficulties: C8D1 (n=111, 43) | 16.8 (25.0) | 15.5 (23.4)
  Financial Difficulties: C9D1 (n=101, 36) | 17.8 (26.1) | 16.7 (23.2)
  Financial Difficulties: C10D1 (n=94, 33) | 16.3 (26.2) | 15.2 (23.7)
  Financial Difficulties: C11D1 (n=84, 25) | 17.5 (25.1) | 17.3 (21.8)
  Financial Difficulties: C12D1 (n=76, 23) | 17.1 (24.6) | 18.8 (28.1)
  Financial Difficulties: C13D1 (n=74, 21) | 16.2 (24.2) | 17.5 (27.1)
  Financial Difficulties: C14D1 (n=66, 19) | 14.1 (20.3) | 17.5 (32.1)
  Financial Difficulties: C15D1 (n=62, 16) | 14.0 (23.0) | 16.7 (27.2)
  Financial Difficulties: C16D1 (n=53, 12) | 15.7 (25.0) | 30.6 (36.1)
  Financial Difficulties: C17D1 (n=47, 11) | 17.7 (29.4) | 33.3 (36.5)
  Financial Difficulties: C18D1 (n=44, 11) | 18.9 (30.0) | 15.2 (31.1)
  Financial Difficulties: C19D1 (n=40, 9) | 17.5 (31.1) | 25.9 (32.4)
  Financial Difficulties: C20D1 (n=35, 8) | 16.2 (27.3) | 25.0 (34.5)
  Financial Difficulties: C21D1 (n=30, 8) | 13.3 (27.1) | 29.2 (33.0)
  Financial Difficulties: C22D1 (n=24, 7) | 18.1 (31.1) | 28.6 (35.6)
  Financial Difficulties: C23D1 (n=23, 4) | 17.4 (31.6) | 33.3 (47.1)
  Financial Difficulties: C24D1 (n=20, 3) | 20.0 (33.2) | 33.3 (57.7)
  Financial Difficulties: C25D1 (n=18, 3) | 11.1 (16.2) | 44.4 (50.9)
  Financial Difficulties: C26D1 (n=14, 3) | 14.3 (17.1) | 44.4 (50.9)
  Financial Difficulties: C27D1 (n=14, 2) | 14.3 (17.1) | 66.7 (47.1)
  Financial Difficulties: C28D1 (n=11, 2) | 15.2 (22.9) | 66.7 (47.1)
  Financial Difficulties: C29D1 (n=8, 2) | 8.3 (15.4) | 66.7 (47.1)
  Financial Difficulties: C30D1 (n=8, 1) | 4.2 (11.8) | 100.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Financial Difficulties: C31D1 (n=7, 0) | 9.5 (16.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Financial Difficulties: C32D1 (n=6, 0) | 22.2 (27.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Financial Difficulties: C33D1 (n=6, 0) | 16.7 (27.9) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Financial Difficulties: C34D1 (n=5, 0) | 13.3 (18.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Financial Difficulties: C35D1 (n=4, 0) | 8.3 (16.7) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Financial Difficulties: C36D1 (n=1, 0) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Financial Difficulties: C37D1 (n=1, 0) | 66.7 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Financial Difficulties: EOT (n=49, 90) | 17.0 (27.3) | 24.1 (30.0)
  Appetite loss: C32D1 (n=6, 0) | 11.1 (17.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Appetite loss: C33D1 (n=6, 0) | 11.1 (17.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Appetite loss: C34D1 (n=5, 0) | 13.3 (18.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Appetite loss: C35D1 (n=4, 0) | 16.7 (19.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Appetite loss: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Appetite loss: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Appetite loss: EOT (n=49, 90) | 21.8 (26.0) | 28.1 (30.4)
  Global Qol: EOT (n=49, 90) | 56.1 (24.5) | 46.4 (25.4)
  Physical Functioning: EOT (n=49, 90) | 80.7 (23.0) | 66.2 (27.7)
  Role Functioning: EOT (n=49, 90) | 71.8 (27.7) | 54.1 (34.7)
  Emotional Functioning: EOT (n=49, 90) | 75.2 (25.1) | 74.5 (25.2)
  Cognitive Functioning: EOT (n=49, 90) | 83.7 (20.3) | 80.0 (24.0)
  Social Function: EOT (n=49, 90) | 78.2 (27.9) | 59.4 (33.5)
  Fatigue: EOT (n=49, 90) | 32.0 (28.2) | 46.9 (26.9)
  Nausea and Vomiting: EOT (n=49, 90) | 16.3 (22.9) | 15.7 (20.4)
  Pain: EOT (n=49, 90) | 23.8 (30.4) | 33.7 (31.3)
  Dyspnea: EOT (n=49, 90) | 23.8 (28.1) | 40.0 (30.1)
  Insomnia: EOT (n=49, 90) | 18.4 (24.6) | 30.4 (27.7)

14. Secondary Outcome: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Supplement Module for Lung Cancer (EORTC QLQ-LC13)
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, chest pain, arm pain, other pain, and medicine for pain). Recall period: past week; response range: 1 'Not at All' to 4 'Very Much'. Scores averaged, transformed to 0-100 scale; higher symptom score = greater degree of symptoms.
Time Frame: Baseline, Day 1 of each cycle until disease progression, end of treatment (up to 112 weeks)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 164 | 162
units on a scale
  Dyspnea: Baseline (n=164, 162) | 27.2 (21.7) | 26.9 (23.4)
  Dyspnea: C2D1 (n=155, 132) | 17.6 (18.1) | 28.6 (22.3)
  Dyspnea: C3D1 (n=153, 106) | 17.9 (17.8) | 28.0 (25.4)
  Dyspnea: C4D1 (n=135, 91) | 16.2 (17.5) | 27.5 (22.8)
  Dyspnea: C5D1 (n=123, 74) | 16.9 (16.7) | 24.8 (22.9)
  Dyspnea: C6D1 (n=119, 70) | 15.2 (15.8) | 25.2 (23.0)
  Dyspnea: C7D1 (n=115, 52) | 15.6 (16.5) | 24.4 (20.3)
  Dyspnea: C8D1 (n=111, 43) | 14.7 (16.0) | 22.0 (22.8)
  Dyspnea: C9D1 (n=101, 37) | 13.9 (15.8) | 19.5 (19.0)
  Dyspnea: C10D1 (n=94, 33) | 15.4 (17.0) | 21.5 (21.0)
  Dyspnea: C11D1 (n=84, 25) | 15.1 (17.5) | 20.4 (24.1)
  Dyspnea: C12D1 (n=76, 23) | 13.7 (15.5) | 22.7 (22.1)
  Dyspnea: C13D1 (n=74, 21) | 12.8 (14.0) | 26.5 (25.9)
  Dyspnea: C14D1 (n=66, 19) | 14.8 (16.9) | 26.3 (26.8)
  Dyspnea: C15D1 (n=62, 16) | 13.2 (15.4) | 22.9 (18.4)
  Dyspnea: C16D1 (n=53, 12) | 12.6 (11.7) | 22.2 (18.3)
  Dyspnea: C17D1 (n=46, 11) | 12.3 (11.5) | 30.3 (23.9)
  Dyspnea: C18D1 (n=45, 11) | 14.1 (13.5) | 26.3 (20.7)
  Dyspnea: C19D1 (n=40, 9) | 14.4 (13.8) | 23.5 (15.2)
  Dyspnea: C20D1 (n=35, 8) | 13.7 (12.9) | 34.7 (24.1)
  Dyspnea: C21D1 (n=30, 8) | 12.6 (13.0) | 25.0 (14.2)
  Dyspnea: C22D1 (n=24, 7) | 10.6 (11.1) | 27.0 (21.1)
  Dyspnea: C23D1 (n=23, 4) | 13.8 (14.2) | 52.8 (19.0)
  Dyspnea: C24D1 (n=20, 3) | 14.4 (14.9) | 48.1 (23.1)
  Dyspnea: C25D1 (n=18, 3) | 15.4 (12.1) | 40.7 (23.1)
  Dyspnea: C26D1 (n=14, 3) | 14.3 (10.2) | 44.4 (22.2)
  Dyspnea: C27D1 (n=14, 2) | 15.1 (11.2) | 55.6 (0.0)
  Dyspnea: C28D1 (n=11, 2) | 11.1 (8.6) | 61.1 (7.9)
  Dyspnea: C29D1 (n=8, 2) | 12.5 (11.0) | 50.0 (7.9)
  Dyspnea: C30D1 (n=8, 1) | 9.7 (7.1) | 77.8 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Dyspnea: C31D1 (n=7, 0) | 15.9 (8.7) | NA (NA) — Data was not analyzed as no participants were evaluable
  Dyspnea: C32D1 (n=6, 0) | 18.5 (9.1) | NA (NA) — Data was not analyzed as no participants were evaluable
  Dyspnea: C33D1 (n=6, 0) | 18.5 (9.1) | NA (NA) — Data was not analyzed as no participants were evaluable
  Dyspnea: C34D1 (n=5, 0) | 20.0 (5.0) | NA (NA) — Data was not analyzed as no participants were evaluable
  Dyspnea: C35D1 (n=4, 0) | 16.7 (6.4) | NA (NA) — Data was not analyzed as no participants were evaluable
  Dyspnea: C36D1 (n=1, 0) | 22.2 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable
  Dyspnea: C37D1 (n=1, 0) | 11.1 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable
  Dyspnea: EOT (n=49, 90) | 21.8 (19.0) | 35.6 (26.7)
  Coughing: Baseline (n=164, 162) | 38.2 (27.4) | 42.2 (31.3)
  Coughing: C2D1 (n=155, 132) | 23.0 (19.6) | 34.8 (26.3)
  Coughing: C3D1 (n=153, 106) | 23.5 (21.6) | 32.4 (27.4)
  Coughing: C4D1 (n=135, 91) | 19.8 (22.4) | 27.1 (24.8)
  Coughing: C5D1 (n=123, 74) | 18.4 (21.0) | 25.7 (25.0)
  Coughing: C6D1 (n=119, 70) | 14.6 (18.2) | 30.0 (25.5)
  Coughing: C7D1 (n=115, 52) | 15.9 (18.4) | 26.3 (23.2)
  Coughing: C8D1 (n=111, 43) | 13.2 (18.7) | 22.5 (23.8)
  Coughing: C9D1 (n=101, 37) | 13.5 (18.4) | 25.2 (28.8)
  Coughing: C10D1 (n=94, 33) | 14.2 (19.2) | 20.2 (26.3)
  Coughing: C11D1 (n=83, 25) | 12.9 (20.7) | 18.7 (25.6)
  Coughing: C12D1 (n=76, 23) | 14.5 (20.6) | 23.2 (25.5)
  Coughing: C13D1 (n=74, 21) | 14.0 (21.4) | 27.0 (27.1)
  Coughing: C14D1 (n=66, 19) | 13.1 (19.3) | 24.6 (31.1)
  Coughing: C15D1 (n=62, 16) | 11.8 (21.0) | 20.8 (20.6)
  Coughing: C16D1 (n=53, 12) | 13.8 (19.0) | 22.2 (21.7)
  Coughing: C17D1 (n=47, 11) | 6.4 (15.0) | 27.3 (25.0)
  Coughing: C18D1 (n=45, 11) | 13.3 (18.0) | 18.2 (17.4)
  Coughing: C19D1 (n=40, 9) | 12.5 (18.0) | 14.8 (17.6)
  Coughing: C20D1 (n=35, 8) | 10.5 (15.7) | 29.2 (21.4)
  Coughing: C21D1 (n=30, 8) | 13.3 (24.1) | 33.3 (25.2)
  Coughing: C22D1 (n=24, 7) | 8.3 (14.7) | 28.6 (23.0)
  Coughing: C23D1 (n=23, 4) | 11.6 (19.1) | 33.3 (0.0)
  Coughing: C24D1 (n=20, 3) | 8.3 (14.8) | 44.4 (19.2)
  Coughing: C25D1 (n=18, 3) | 5.6 (12.8) | 44.4 (19.2)
  Coughing: C26D1 (n=14, 3) | 2.4 (8.9) | 33.3 (0.0)
  Coughing: C27D1 (n=14, 2) | 7.1 (14.2) | 50.0 (23.6)
  Coughing: C28D1 (n=11, 2) | 18.2 (31.1) | 50.0 (23.6)
  Coughing: C29D1 (n=8, 2) | 8.3 (15.4) | 33.3 (0.0)
  Coughing: C30D1 (n=8, 1) | 20.8 (24.8) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Coughing: C31D1 (n=7, 0) | 19.0 (17.8) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Coughing: C32D1 (n=6, 0) | 16.7 (27.9) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Coughing: C33D1 (n=6, 0) | 11.1 (17.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Coughing: C34D1 (n=5, 0) | 20.0 (29.8) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Coughing: C35D1 (n=4, 0) | 33.3 (47.1) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Coughing: C36D1 (n=1, 0) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Coughing: C37D1 (n=1, 0) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Coughing: EOT (n=49, 90) | 25.9 (23.8) | 37.4 (29.1)
  Hemoptysis: Baseline (n=164, 162) | 2.4 (9.5) | 3.7 (12.3)
  Hemoptysis: C2D1 (n=155, 132) | 1.7 (7.4) | 3.5 (12.5)
  Hemoptysis: C3D1 (n=153, 106) | 0.9 (5.3) | 2.2 (8.3)
  Hemoptysis: C4D1 (n=135, 91) | 1.0 (5.7) | 1.5 (6.9)
  Hemoptysis: C5D1 (n=123, 74) | 0.3 (3.0) | 0.9 (5.4)
  Hemoptysis: C6D1 (n=119, 70) | 0.6 (4.3) | 3.8 (14.5)
  Hemoptysis: C7D1 (n=115, 52) | 0.0 (0.0) | 1.3 (9.2)
  Hemoptysis: C8D1 (n=111, 43) | 0.9 (7.0) | 2.3 (11.3)
  Hemoptysis: C9D1 (n=101, 37) | 0.3 (3.3) | 2.7 (12.1)
  Hemoptysis: C10D1 (n=94, 33) | 0.4 (3.4) | 3.0 (17.4)
  Hemoptysis: C11D1 (n=83, 25) | 2.4 (11.4) | 4.0 (14.7)
  Hemoptysis: C12D1 (n=76, 23) | 0.9 (5.4) | 5.8 (21.7)
  Hemoptysis: C13D1 (n=74, 21) | 2.3 (10.1) | 4.8 (15.9)
  Hemoptysis: C14D1 (n=66, 19) | 0.5 (4.1) | 0.0 (0.0)
  Hemoptysis: C15D1 (n=62, 16) | 1.1 (5.9) | 0.0 (0.0)
  Hemoptysis: C16D1 (n=53, 12) | 0.6 (4.6) | 5.6 (13.0)
  Hemoptysis: C17D1 (n=47, 11) | 0.0 (0.0) | 9.1 (21.6)
  Hemoptysis: C18D1 (n=45, 11) | 1.5 (6.9) | 3.0 (10.1)
  Hemoptysis: C19D1 (n=40, 9) | 0.0 (0.0) | 3.7 (11.1)
  Hemoptysis: C20D1 (n=35, 8) | 1.0 (5.6) | 8.3 (15.4)
  Hemoptysis: C21D1 (n=30, 8) | 0.0 (0.0) | 4.2 (11.8)
  Hemoptysis: C22D1 (n=24, 7) | 0.0 (0.0) | 9.5 (16.3)
  Hemoptysis: C23D1 (n=23, 4) | 1.4 (7.0) | 0.0 (0.0)
  Hemoptysis: C24D1 (n=20, 3) | 0.0 (0.0) | 0.0 (0.0)
  Hemoptysis: C25D1 (n=18, 3) | 0.0 (0.0) | 0.0 (0.0)
  Hemoptysis: C26D1 (n=14, 3) | 0.0 (0.0) | 0.0 (0.0)
  Hemoptysis: C27D1 (n=14, 2) | 0.0 (0.0) | 0.0 (0.0)
  Hemoptysis: C28D1 (n=11, 2) | 0.0 (0.0) | 0.0 (0.0)
  Hemoptysis: C29D1 (n=8, 2) | 0.0 (0.0) | 0.0 (0.0)
  Hemoptysis: C30D1 (n=8, 1) | 0.0 (0.0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Hemoptysis: C31D1 (n=7, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Hemoptysis: C32D1 (n=6, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Hemoptysis: C33D1 (n=6, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Hemoptysis: C34D1 (n=5, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Hemoptysis: C35D1 (n=4, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Hemoptysis: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Hemoptysis: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Hemoptysis: EOT (n=49, 90) | 0.7 (4.8) | 4.8 (13.7)
  Sore Mouth: Baseline (n=164, 162) | 5.5 (15.3) | 6.4 (18.4)
  Sore Mouth: C2D1 (n=155, 132) | 8.0 (17.9) | 9.1 (18.5)
  Sore Mouth: C3D1 (n=153, 106) | 7.0 (14.6) | 9.4 (21.0)
  Sore Mouth: C4D1 (n=135, 91) | 8.1 (16.5) | 10.3 (21.5)
  Sore Mouth: C5D1 (n=123, 73) | 5.1 (12.1) | 9.6 (20.4)
  Sore Mouth: C6D1 (n=119, 70) | 4.8 (13.9) | 10.5 (19.3)
  Sore Mouth: C7D1 (n=115, 52) | 5.2 (15.0) | 7.7 (15.6)
  Sore Mouth: C8D1 (n=111, 43) | 3.0 (9.6) | 10.9 (18.9)
  Sore Mouth: C9D1 (n=101, 37) | 4.8 (12.5) | 10.8 (22.3)
  Sore Mouth: C10D1 (n=94, 33) | 6.4 (14.9) | 12.1 (23.3)
  Sore Mouth: C11D1 (n=84, 25) | 4.8 (14.8) | 9.3 (18.1)
  Sore Mouth: C12D1 (n=76, 23) | 3.9 (12.1) | 8.7 (18.0)
  Sore Mouth: C13D1 (n=74, 21) | 4.5 (12.7) | 9.5 (15.4)
  Sore Mouth: C14D1 (n=66, 19) | 4.5 (12.9) | 7.0 (14.0)
  Sore Mouth: C15D1 (n=62, 16) | 5.4 (12.4) | 14.6 (29.7)
  Sore Mouth: C16D1 (n=53, 12) | 6.3 (14.7) | 8.3 (15.1)
  Sore Mouth: C17D1 (n=47, 11) | 3.5 (10.4) | 6.1 (13.5)
  Sore Mouth: C18D1 (n=45, 11) | 5.2 (12.2) | 12.1 (16.8)
  Sore Mouth: C19D1 (n=40, 9) | 4.2 (11.2) | 7.4 (14.7)
  Sore Mouth: C20D1 (n=35, 8) | 7.6 (16.3) | 12.5 (24.8)
  Sore Mouth: C21D1 (n=30, 8) | 4.4 (11.5) | 4.2 (11.8)
  Sore Mouth: C22D1 (n=24, 7) | 5.6 (12.7) | 7.1 (13.1)
  Sore Mouth: C23D1 (n=23, 4) | 5.1 (11.7) | 16.7 (19.2)
  Sore Mouth: C24D1 (n=20, 3) | 6.7 (17.4) | 0.0 (0.0)
  Sore Mouth: C25D1 (n=18, 3) | 0.0 (0.0) | 0.0 (0.0)
  Sore Mouth: C26D1 (n=14, 3) | 4.8 (17.8) | 11.1 (19.2)
  Sore Mouth: C27D1 (n=14, 2) | 7.1 (19.3) | 16.7 (23.6)
  Sore Mouth: C28D1 (n=11, 2) | 6.1 (20.1) | 0.0 (0.0)
  Sore Mouth: C29D1 (n=8, 2) | 8.3 (15.4) | 16.7 (23.6)
  Sore Mouth: C30D1 (n=8, 1) | 8.3 (23.6) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Sore Mouth: C31D1 (n=7, 0) | 9.5 (25.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Sore Mouth: C32D1 (n=6, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Sore Mouth: C33D1 (n=6, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Sore Mouth: C34D1 (n=5, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Sore Mouth: C35D1 (n=4, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Sore Mouth: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Sore Mouth: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Sore Mouth: EOT (n=49, 90) | 3.4 (10.2) | 8.1 (18.2)
  Dysphagia: Baseline (n=164, 162) | 7.1 (16.4) | 8.6 (20.9)
  Dysphagia: C2D1 (n=155, 132) | 8.2 (15.4) | 9.8 (19.2)
  Dysphagia: C3D1 (n=153, 106) | 7.6 (16.4) | 9.7 (20.6)
  Dysphagia: C4D1 (n=135, 91) | 6.2 (15.3) | 8.1 (19.5)
  Dysphagia: C5D1 (n=123, 74) | 6.0 (14.8) | 7.7 (17.0)
  Dysphagia: C6D1 (n=119, 70) | 7.0 (15.0) | 10.0 (16.4)
  Dysphagia: C7D1 (n=115, 52) | 4.1 (11.8) | 5.1 (13.8)
  Dysphagia: C8D1 (n=111, 43) | 3.2 (11.1) | 6.2 (15.0)
  Dysphagia: C9D1 (n=101, 37) | 5.0 (11.9) | 7.2 (16.0)
  Dysphagia: C10D1 (n=94, 33) | 4.3 (12.2) | 6.1 (13.1)
  Dysphagia: C11D1 (n=84, 25) | 3.2 (9.8) | 4.0 (11.1)
  Dysphagia: C12D1 (n=76, 23) | 3.5 (10.3) | 7.2 (17.3)
  Dysphagia: C13D1 (n=74, 21) | 4.1 (11.0) | 6.3 (13.4)
  Dysphagia: C14D1 (n=66, 19) | 3.0 (11.3) | 7.0 (14.0)
  Dysphagia: C15D1 (n=62, 16) | 3.8 (13.6) | 4.2 (16.7)
  Dysphagia: C16D1 (n=53, 12) | 4.4 (11.4) | 2.8 (9.6)
  Dysphagia: C17D1 (n=47, 11) | 2.8 (9.4) | 6.1 (13.5)
  Dysphagia: C18D1 (n=45, 11) | 3.7 (10.6) | 3.0 (10.1)
  Dysphagia: C19D1 (n=40, 9) | 4.2 (11.2) | 0.0 (0.0)
  Dysphagia: C20D1 (n=35, 8) | 4.8 (14.3) | 8.3 (15.4)
  Dysphagia: C21D1 (n=30, 8) | 3.3 (10.2) | 8.3 (15.4)
  Dysphagia: C22D1 (n=24, 7) | 2.8 (9.4) | 0.0 (0.0)
  Dysphagia: C23D1 (n=23, 4) | 2.9 (9.6) | 8.3 (16.7)
  Dysphagia: C24D1 (n=20, 3) | 5.0 (22.4) | 0.0 (0.0)
  Dysphagia: C25D1 (n=18, 3) | 0.0 (0.0) | 11.1 (19.2)
  Dysphagia: C26D1 (n=14, 3) | 9.5 (27.5) | 11.1 (19.2)
  Dysphagia: C27D1 (n=14, 2) | 2.4 (8.9) | 16.7 (23.6)
  Dysphagia: C28D1 (n=11, 2) | 6.1 (13.5) | 16.7 (23.6)
  Dysphagia: C29D1 (n=8, 2) | 8.3 (15.4) | 16.7 (23.6)
  Dysphagia: C30D1 (n=8, 1) | 0.0 (0.0) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Dysphagia: C31D1 (n=7, 0) | 4.8 (12.6) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dysphagia: C32D1 (n=6, 0) | 5.6 (13.6) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dysphagia: C33D1 (n=6, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dysphagia: C34D1 (n=5, 0) | 6.7 (14.9) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dysphagia: C35D1 (n=4, 0) | 8.3 (16.7) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dysphagia: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dysphagia: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Dysphagia: EOT (n=49, 90) | 4.8 (13.6) | 8.5 (19.7)
  Peripheral Neuropathy: Baseline (n=164, 162) | 14.0 (22.1) | 17.7 (27.3)
  Peripheral Neuropathy: C2D1 (n=155, 132) | 18.1 (24.1) | 21.5 (29.2)
  Peripheral Neuropathy: C3D1 (n=153, 106) | 17.6 (26.2) | 18.2 (29.1)
  Peripheral Neuropathy: C4D1 (n=134, 91) | 15.9 (23.0) | 21.6 (27.8)
  Peripheral Neuropathy: C5D1 (n=123, 74) | 15.2 (21.0) | 21.2 (28.4)
  Peripheral Neuropathy: C6D1 (n=119, 70) | 13.7 (21.9) | 18.1 (27.0)
  Peripheral Neuropathy: C7D1 (n=115, 52) | 13.0 (21.0) | 21.8 (28.7)
  Peripheral Neuropathy: C8D1 (n=111, 43) | 10.8 (20.2) | 24.0 (32.8)
  Peripheral Neuropathy: C9D1 (n=101, 37) | 11.2 (19.6) | 29.7 (34.1)
  Peripheral Neuropathy: C10D1 (n=94, 33) | 11.3 (21.1) | 27.3 (29.4)
  Peripheral Neuropathy: C11D1 (n=84, 25) | 11.1 (21.5) | 24.0 (31.2)
  Peripheral Neuropathy: C12D1 (n=76, 23) | 11.4 (22.1) | 33.3 (36.2)
  Peripheral Neuropathy: C13D1 (n=74, 21) | 10.4 (19.1) | 33.3 (35.0)
  Peripheral Neuropathy: C14D1 (n=66, 19) | 10.6 (21.2) | 29.8 (35.0)
  Peripheral Neuropathy: C15D1 (n=62, 16) | 8.6 (18.0) | 25.0 (31.0)
  Peripheral Neuropathy: C16D1 (n=52, 12) | 10.3 (19.3) | 25.0 (20.7)
  Peripheral Neuropathy: C17D1 (n=47, 11) | 12.1 (23.5) | 27.3 (29.1)
  Peripheral Neuropathy: C18D1 (n=45, 11) | 11.9 (22.6) | 30.3 (31.5)
  Peripheral Neuropathy: C19D1 (n=40, 9) | 9.2 (20.0) | 22.2 (16.7)
  Peripheral Neuropathy: C20D1 (n=35, 8) | 12.4 (25.7) | 33.3 (30.9)
  Peripheral Neuropathy: C21D1 (n=30, 8) | 11.1 (18.2) | 29.2 (21.4)
  Peripheral Neuropathy: C22D1 (n=24, 7) | 8.3 (20.3) | 28.6 (23.0)
  Peripheral Neuropathy: C23D1 (n=23, 4) | 8.7 (20.6) | 41.7 (31.9)
  Peripheral Neuropathy: C24D1 (n=20, 3) | 3.3 (14.9) | 44.4 (38.5)
  Peripheral Neuropathy: C25D1 (n=18, 3) | 9.3 (19.2) | 44.4 (38.5)
  Peripheral Neuropathy: C26D1 (n=14, 3) | 16.7 (36.4) | 22.2 (19.2)
  Peripheral Neuropathy: C27D1 (n=14, 2) | 9.5 (20.4) | 66.7 (0.0)
  Peripheral Neuropathy: C28D1 (n=11, 2) | 15.2 (22.9) | 33.3 (0.0)
  Peripheral Neuropathy: C29D1 (n=8, 2) | 12.5 (24.8) | 50.0 (23.6)
  Peripheral Neuropathy: C30D1 (n=8, 1) | 16.7 (30.9) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Peripheral Neuropathy: C31D1 (n=7, 0) | 19.0 (32.5) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Peripheral Neuropathy: C32D1 (n=6, 0) | 11.1 (27.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Peripheral Neuropathy: C33D1 (n=6, 0) | 11.1 (27.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Peripheral Neuropathy: C34D1 (n=5, 0) | 20.0 (44.7) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Peripheral Neuropathy: C35D1 (n=4, 0) | 25.0 (50.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Peripheral Neuropathy: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Peripheral Neuropathy: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Peripheral Neuropathy: EOT (n=49, 90) | 10.2 (16.9) | 21.9 (29.6)
  Alopecia: Baseline (n=163, 162) | 17.4 (30.6) | 16.9 (29.8)
  Alopecia: C2D1 (n=155, 132) | 9.5 (21.4) | 36.6 (39.7)
  Alopecia: C3D1 (n=153, 106) | 7.6 (18.1) | 30.5 (36.5)
  Alopecia: C4D1 (n=135, 91) | 8.9 (22.0) | 24.9 (32.0)
  Alopecia: C5D1 (n=123, 74) | 6.0 (17.1) | 23.9 (31.0)
  Alopecia: C6D1 (n=118, 70) | 4.2 (14.8) | 23.3 (32.8)
  Alopecia: C7D1 (n=115, 52) | 4.9 (14.1) | 19.9 (30.4)
  Alopecia: C8D1 (n=111, 43) | 3.9 (11.7) | 18.6 (28.5)
  Alopecia: C9D1 (n=101, 37) | 4.0 (11.8) | 16.2 (23.1)
  Alopecia: C10D1 (n=94, 33) | 4.6 (14.3) | 14.1 (22.1)
  Alopecia: C11D1 (n=84, 25) | 4.0 (15.0) | 16.0 (21.8)
  Alopecia: C12D1 (n=76, 23) | 4.4 (14.7) | 20.3 (26.1)
  Alopecia: C13D1 (n=74, 21) | 6.3 (18.0) | 12.7 (19.7)
  Alopecia: C14D1 (n=65, 19) | 3.6 (14.6) | 15.8 (23.2)
  Alopecia: C15D1 (n=62, 16) | 4.8 (16.9) | 8.3 (19.2)
  Alopecia: C16D1 (n=53, 12) | 6.3 (18.6) | 13.9 (22.3)
  Alopecia: C17D1 (n=46, 11) | 5.1 (17.2) | 18.2 (22.9)
  Alopecia: C18D1 (n=45, 11) | 3.7 (12.8) | 18.2 (22.9)
  Alopecia: C19D1 (n=40, 9) | 5.8 (19.8) | 18.5 (24.2)
  Alopecia: C20D1 (n=35, 8) | 3.8 (13.5) | 25.0 (23.6)
  Alopecia: C21D1 (n=30, 8) | 7.8 (22.6) | 16.7 (25.2)
  Alopecia: C22D1 (n=24, 7) | 2.8 (9.4) | 14.3 (17.8)
  Alopecia: C23D1 (n=23, 3) | 1.4 (7.0) | 22.2 (19.2)
  Alopecia: C24D1 (n=20, 3) | 6.7 (23.2) | 33.3 (33.3)
  Alopecia: C25D1 (n=18, 3) | 9.3 (27.5) | 33.3 (33.3)
  Alopecia: C26D1 (n=14, 3) | 7.1 (26.7) | 44.4 (38.5)
  Alopecia: C27D1 (n=14, 2) | 16.7 (36.4) | 33.3 (0.0)
  Alopecia: C28D1 (n=11, 2) | 6.1 (20.1) | 50.0 (23.6)
  Alopecia: C29D1 (n=8, 2) | 16.7 (35.6) | 33.3 (0.0)
  Alopecia: C30D1 (n=8, 1) | 12.5 (35.4) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Alopecia: C31D1 (n=7, 0) | 9.5 (25.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Alopecia: C32D1 (n=6, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Alopecia: C33D1 (n=6, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Alopecia: C34D1 (n=5, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Alopecia: C35D1 (n=4, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Alopecia: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Alopecia: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Alopecia: EOT (n=49, 90) | 6.8 (18.0) | 33.3 (37.7)
  Pain in Chest: Baseline (n=163, 160) | 18.8 (22.8) | 24.0 (27.5)
  Pain in Chest: C2D1 (n=155, 132) | 9.5 (17.7) | 23.7 (25.9)
  Pain in Chest: C3D1 (n=153, 106) | 7.0 (13.6) | 23.3 (26.5)
  Pain in Chest: C4D1 (n=135, 91) | 7.4 (13.9) | 19.8 (22.8)
  Pain in Chest: C5D1 (n=123, 74) | 6.8 (14.1) | 17.1 (21.5)
  Pain in Chest: C6D1 (n=119, 70) | 6.2 (13.0) | 16.2 (22.5)
  Pain in Chest: C7D1 (n=115, 52) | 7.5 (14.7) | 16.7 (22.4)
  Pain in Chest: C8D1 (n=111, 43) | 5.1 (14.4) | 14.0 (20.9)
  Pain in Chest: C9D1 (n=101, 37) | 5.9 (12.8) | 17.1 (23.1)
  Pain in Chest: C10D1 (n=94, 33) | 6.7 (14.3) | 18.2 (31.3)
  Pain in Chest: C11D1 (n=84, 25) | 6.3 (13.2) | 20.0 (25.5)
  Pain in Chest: C12D1 (n=76, 23) | 5.3 (12.2) | 23.2 (30.9)
  Pain in Chest: C13D1 (n=74, 21) | 6.3 (13.1) | 23.8 (30.1)
  Pain in Chest: C14D1 (n=66, 19) | 7.6 (16.3) | 22.8 (22.4)
  Pain in Chest: C15D1 (n=62, 16) | 5.9 (14.2) | 18.7 (24.2)
  Pain in Chest: C16D1 (n=53, 12) | 3.8 (10.7) | 16.7 (17.4)
  Pain in Chest: C17D1 (n=46, 11) | 7.2 (15.6) | 21.2 (22.5)
  Pain in Chest: C18D1 (n=45, 11) | 5.9 (16.3) | 24.2 (33.6)
  Pain in Chest: C19D1 (n=40, 9) | 5.0 (14.2) | 18.5 (24.2)
  Pain in Chest: C20D1 (n=35, 8) | 5.7 (15.1) | 29.2 (21.4)
  Pain in Chest: C21D1 (n=30, 8) | 5.6 (15.4) | 25.0 (23.6)
  Pain in Chest: C22D1 (n=24, 7) | 4.2 (11.3) | 26.2 (30.2)
  Pain in Chest: C23D1 (n=23, 4) | 3.6 (10.0) | 41.7 (31.9)
  Pain in Chest: C24D1 (n=20, 3) | 1.7 (7.5) | 33.3 (33.3)
  Pain in Chest: C25D1 (n=18, 3) | 5.6 (12.8) | 33.3 (33.3)
  Pain in Chest: C26D1 (n=14, 3) | 7.1 (19.3) | 33.3 (33.3)
  Pain in Chest: C27D1 (n=14, 2) | 4.8 (12.1) | 50.0 (23.6)
  Pain in Chest: C28D1 (n=11, 2) | 9.1 (15.6) | 50.0 (23.6)
  Pain in Chest: C29D1 (n=8, 2) | 0.0 (0.0) | 50.0 (23.6)
  Pain in Chest: C30D1 (n=8, 1) | 4.2 (11.8) | 66.7 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pain in Chest: C31D1 (n=7, 0) | 9.5 (16.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Chest: C32D1 (n=6, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Chest: C33D1 (n=6, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Chest: C34D1 (n=5, 0) | 6.7 (14.9) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Chest: C35D1 (n=4, 0) | 8.3 (16.7) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Chest: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Chest: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Chest: EOT (n=49, 90) | 17.0 (24.6) | 28.5 (29.4)
  Pain in Arm or Shoulder: Baseline (n=164, 161) | 16.3 (24.1) | 19.5 (28.0)
  Pain in Arm or Shoulder: C2D1 (n=155, 132) | 9.0 (18.3) | 19.9 (27.0)
  Pain in Arm or Shoulder: C3D1 (n=153, 105) | 8.1 (14.8) | 17.5 (24.5)
  Pain in Arm or Shoulder: C4D1 (n=135, 91) | 6.9 (15.3) | 14.3 (22.3)
  Pain in Arm or Shoulder: C5D1 (n=123, 74) | 6.2 (15.0) | 13.1 (21.9)
  Pain in Arm or Shoulder: C6D1 (n=119, 70) | 6.7 (14.1) | 17.1 (25.8)
  Pain in Arm or Shoulder: C7D1 (n=115, 52) | 6.4 (13.2) | 17.3 (23.3)
  Pain in Arm or Shoulder: C8D1 (n=111, 43) | 6.9 (14.3) | 20.2 (28.3)
  Pain in Arm or Shoulder: C9D1 (n=101, 37) | 5.6 (12.5) | 23.4 (28.2)
  Pain in Arm or Shoulder: C10D1 (n=94, 33) | 7.4 (17.0) | 25.3 (32.3)
  Pain in Arm or Shoulder: C11D1 (n=84, 25) | 6.0 (14.8) | 24.0 (26.4)
  Pain in Arm or Shoulder: C12D1 (n=76, 23) | 6.6 (15.4) | 29.0 (35.3)
  Pain in Arm or Shoulder: C13D1 (n=74, 21) | 5.9 (12.8) | 25.4 (34.8)
  Pain in Arm or Shoulder: C14D1 (n=66, 19) | 7.6 (18.3) | 29.8 (31.2)
  Pain in Arm or Shoulder: C15D1 (n=62, 16) | 5.4 (13.8) | 25.0 (25.8)
  Pain in Arm or Shoulder: C16D1 (n=53, 12) | 5.0 (12.0) | 16.7 (22.5)
  Pain in Arm or Shoulder: C17D1 (n=47, 11) | 3.5 (10.4) | 21.2 (22.5)
  Pain in Arm or Shoulder: C18D1 (n=45, 11) | 8.1 (20.3) | 30.3 (34.8)
  Pain in Arm or Shoulder: C19D1 (n=40, 9) | 6.7 (15.5) | 18.5 (24.2)
  Pain in Arm or Shoulder: C20D1 (n=35, 8) | 9.5 (22.2) | 25.0 (23.6)
  Pain in Arm or Shoulder: C21D1 (n=30, 8) | 7.8 (16.8) | 29.2 (27.8)
  Pain in Arm or Shoulder: C22D1 (n=24, 7) | 2.8 (9.4) | 21.4 (24.9)
  Pain in Arm or Shoulder: C23D1 (n=23, 4) | 0.7 (3.5) | 33.3 (38.5)
  Pain in Arm or Shoulder: C24D1 (n=20, 3) | 3.3 (10.3) | 44.4 (38.5)
  Pain in Arm or Shoulder: C25D1 (n=18, 3) | 1.9 (7.9) | 33.3 (33.3)
  Pain in Arm or Shoulder: C26D1 (n=14, 3) | 7.1 (19.3) | 22.2 (19.2)
  Pain in Arm or Shoulder: C27D1 (n=14, 2) | 4.8 (12.1) | 50.0 (23.6)
  Pain in Arm or Shoulder: C28D1 (n=11, 2) | 0.0 (0.0) | 33.3 (0.0)
  Pain in Arm or Shoulder: C29D1 (n=8, 2) | 0.0 (0.0) | 66.7 (0.0)
  Pain in Arm or Shoulder: C30D1 (n=8, 1) | 0.0 (0.0) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pain in Arm or Shoulder: C31D1 (n=7, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Arm or Shoulder: C32D1 (n=6, 0) | 11.1 (17.2) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Arm or Shoulder: C33D1 (n=6, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Arm or Shoulder: C34D1 (n=5, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Arm or Shoulder: C35D1 (n=4, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Arm or Shoulder: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Arm or Shoulder: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Arm or Shoulder: EOT (n=48, 90) | 11.1 (21.0) | 21.9 (28.8)
  Pain in Other Parts: Baseline (n=163, 158) | 23.1 (27.3) | 31.4 (30.4)
  Pain in Other Parts: C2D1 (n=153, 125) | 15.0 (23.2) | 25.9 (28.0)
  Pain in Other Parts: C3D1 (n=152, 104) | 11.4 (20.7) | 21.2 (27.1)
  Pain in Other Parts: C4D1 (n=134, 90) | 12.7 (22.7) | 21.5 (24.6)
  Pain in Other Parts: C5D1 (n=123, 73) | 14.4 (23.0) | 20.5 (27.6)
  Pain in Other Parts: C6D1 (n=118, 68) | 10.7 (18.9) | 18.1 (26.0)
  Pain in Other Parts: C7D1 (n=115, 51) | 11.3 (20.7) | 16.3 (26.1)
  Pain in Other Parts: C8D1 (n=111, 42) | 10.5 (20.6) | 22.2 (30.9)
  Pain in Other Parts: C9D1 (n=100, 37) | 10.7 (21.1) | 24.3 (31.1)
  Pain in Other Parts: C10D1 (n=92, 33) | 9.8 (18.8) | 28.3 (35.5)
  Pain in Other Parts: C11D1 (n=83, 25) | 12.4 (21.3) | 24.0 (29.7)
  Pain in Other Parts: C12D1 (n=74, 23) | 12.2 (20.3) | 24.6 (30.5)
  Pain in Other Parts: C13D1 (n=74, 21) | 10.8 (19.2) | 31.7 (34.1)
  Pain in Other Parts: C14D1 (n=66, 19) | 11.6 (18.0) | 24.6 (29.1)
  Pain in Other Parts: C15D1 (n=61, 16) | 9.8 (15.3) | 25.0 (22.8)
  Pain in Other Parts: C16D1 (n=53, 12) | 10.7 (19.4) | 38.9 (34.3)
  Pain in Other Parts: C17D1 (n=46, 11) | 13.8 (19.3) | 24.2 (21.6)
  Pain in Other Parts: C18D1 (n=45, 11) | 10.4 (19.9) | 33.3 (39.4)
  Pain in Other Parts: C19D1 (n=40, 9) | 14.2 (22.5) | 25.9 (14.7)
  Pain in Other Parts: C20D1 (n=35, 8) | 13.3 (20.1) | 29.2 (21.4)
  Pain in Other Parts: C21D1 (n=30, 8) | 21.1 (27.0) | 29.2 (37.5)
  Pain in Other Parts: C22D1 (n=24, 7) | 12.5 (21.6) | 40.5 (30.2)
  Pain in Other Parts: C23D1 (n=23, 4) | 5.1 (11.7) | 41.7 (31.9)
  Pain in Other Parts: C24D1 (n=20, 3) | 6.7 (17.4) | 11.1 (19.2)
  Pain in Other Parts: C25D1 (n=18, 3) | 9.3 (15.4) | 44.4 (38.5)
  Pain in Other Parts: C26D1 (n=14, 3) | 23.8 (30.5) | 33.3 (33.3)
  Pain in Other Parts: C27D1 (n=14, 2) | 16.7 (31.4) | 50.0 (23.6)
  Pain in Other Parts: C28D1 (n=11, 2) | 6.1 (13.5) | 33.3 (0.0)
  Pain in Other Parts: C29D1 (n=8, 2) | 4.2 (11.8) | 16.7 (23.6)
  Pain in Other Parts: C30D1 (n=8, 1) | 12.5 (17.3) | 33.3 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Pain in Other Parts: C31D1 (n=7, 0) | 9.5 (16.3) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Other Parts: C32D1 (n=6, 0) | 5.6 (13.6) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Other Parts: C33D1 (n=6, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Other Parts: C34D1 (n=5, 0) | 6.7 (14.9) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Other Parts: C35D1 (n=4, 0) | 0.0 (0.0) | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Other Parts: C36D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Other Parts: C37D1 (n=1, 0) | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Pain in Other Parts: EOT (n=49, 90) | 18.4 (29.7) | 29.6 (34.8)

15. Secondary Outcome: European Quality of Life - 5 Dimensional (EQ-5D) Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Day 1 of each cycle until disease progression, end of treatment (up to 112 weeks)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Crizotinib | Chemotherapy
Number analyzed (Participants) | 164 | 161
units on a scale
  Baseline (n=164, 161) | 64.09 (21.04) | 66.76 (20.74)
  C2D1 (n=153, 131) | 69.19 (19.42) | 66.33 (20.30)
  C3D1 (n=153, 105) | 73.13 (18.97) | 65.84 (20.80)
  C4D1 (n=135, 90) | 73.78 (18.25) | 69.13 (18.14)
  C5D1 (n=122, 74) | 75.27 (17.99) | 68.12 (23.19)
  C6D1 (n=120, 70) | 75.79 (18.67) | 69.71 (22.46)
  C7D1 (n=115, 52) | 77.02 (17.34) | 70.63 (24.31)
  C8D1 (n=110, 43) | 74.72 (18.09) | 72.30 (23.54)
  C9D1 (n=101, 37) | 74.45 (18.32) | 72.27 (25.85)
  C10D1 (n=94, 33) | 75.49 (18.18) | 74.27 (24.88)
  C11D1 (n=84, 25) | 76.32 (17.00) | 77.24 (20.31)
  C12D1 (n=77, 23) | 76.95 (17.63) | 74.83 (22.60)
  C13D1 (n=73, 21) | 76.38 (17.50) | 73.00 (23.54)
  C14D1 (n=66, 19) | 78.77 (15.54) | 74.11 (22.56)
  C15D1 (n=62, 16) | 77.71 (16.78) | 77.44 (19.52)
  C16D1 (n=53, 12) | 75.32 (16.21) | 79.00 (13.28)
  C17D1 (n=47, 11) | 75.09 (17.68) | 81.73 (15.98)
  C18D1 (n=45, 11) | 75.87 (16.63) | 78.91 (16.25)
  C19D1 (n=40, 9) | 76.85 (16.39) | 78.00 (14.04)
  C20D1 (n=35, 8) | 72.66 (19.81) | 76.75 (17.65)
  C21D1 (n=30, 8) | 74.13 (16.19) | 73.63 (19.41)
  C22D1 (n=24, 7) | 77.54 (17.54) | 72.21 (19.79)
  C23D1 (n=23, 4) | 75.48 (17.75) | 54.00 (16.35)
  C24D1 (n=20, 3) | 71.40 (23.15) | 62.00 (20.30)
  C25D1 (n=18, 3) | 75.61 (15.97) | 63.67 (22.59)
  C26D1 (n=14, 3) | 72.14 (20.71) | 63.00 (17.52)
  C27D1 (n=14, 2) | 66.57 (16.96) | 50.00 (14.14)
  C28D1 (n=11, 2) | 72.36 (12.72) | 55.00 (21.21)
  C29D1 (n=8, 2) | 71.38 (12.28) | 45.00 (14.14)
  C30D1 (n=8, 1) | 69.50 (17.00) | 40.00 (NA) — Standard deviation was not estimable since only one participant was evaluable
  C31D1 (n=7, 0) | 68.57 (16.76) | NA (NA) — Data was not analyzed as no participants were evaluable
  C32D1 (n=6, 0) | 65.83 (19.41) | NA (NA) — Data was not analyzed as no participants were evaluable
  C33D1 (n=6, 0) | 67.50 (20.34) | NA (NA) — Data was not analyzed as no participants were evaluable
  C34D1 (n=5, 0) | 68.00 (20.80) | NA (NA) — Data was not analyzed as no participants were evaluable
  C35D1 (n=4, 0) | 72.25 (14.84) | NA (NA) — Data was not analyzed as no participants were evaluable
  C36D1 (n=1, 0) | 90.00 (NA) — Standard deviation was not estimable since only one participant was evaluable | NA (NA) — Data was not analyzed as no participants were evaluable
  C37D1 (n=1, 0) | 85.00 (NA) — Standard deviation was not estimable since only one participant was evaluable | NA (NA) — Data was not analyzed as no participants were evaluable
  EOT (n=49, 90) | 68.33 (21.25) | 58.34 (23.71)

ADVERSE EVENTS:
Time Frame: Active reporting period is from the time of informed consent until at least 28 days after the last dose of study treatment.
Description: All causality (serious and non-serious) adverse events have been reported. Non-serious adverse events above the 5% threshold are reported herein.
Arm/Group | Crizotinib | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 80/172 | 42/171
Other Adverse Events (participants affected / at risk) | 172/172 | 169/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib (N=172) | Chemotherapy (N=171)
Product contamination microbial (General disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 12
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Chest pain (General disorders) | 0 | 2
Death (General disorders) | 2 | 0
Disease progression (General disorders) | 18 | 3
Fatigue (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 1
Sudden death (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Lung abscess (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 8 | 3
Pneumonia bacterial (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood glucose increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Haemoglobin (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Intracranial pressure increased (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Cancer surgery (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Syncope (Cardiac disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral cyst (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 1
Delirium (Psychiatric disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib (N=172) | Chemotherapy (N=171)
Anaemia (Blood and lymphatic system disorders) | 36 | 27
Leukopenia (Blood and lymphatic system disorders) | 24 | 9
Photopsia (Eye disorders) | 21 | 1
Vision blurred (Eye disorders) | 13 | 5
Visual impairment (Eye disorders) | 74 | 8
Abdominal pain (Gastrointestinal disorders) | 18 | 8
Abdominal pain upper (Gastrointestinal disorders) | 17 | 13
Constipation (Gastrointestinal disorders) | 83 | 39
Diarrhoea (Gastrointestinal disorders) | 106 | 34
Dyspepsia (Gastrointestinal disorders) | 18 | 6
Nausea (Gastrointestinal disorders) | 104 | 60
Stomatitis (Gastrointestinal disorders) | 9 | 13
Vomiting (Gastrointestinal disorders) | 88 | 32
Asthenia (General disorders) | 31 | 32
Chest pain (General disorders) | 15 | 13
Fatigue (General disorders) | 51 | 60
Oedema (General disorders) | 15 | 6
Oedema peripheral (General disorders) | 59 | 15
Pyrexia (General disorders) | 41 | 33
Nasopharyngitis (Infections and infestations) | 32 | 7
Upper respiratory tract infection (Infections and infestations) | 24 | 14
Alanine aminotransferase increased (Investigations) | 72 | 21
Aspartate aminotransferase increased (Investigations) | 55 | 17
Blood alkaline phosphatase increased (Investigations) | 18 | 6
Blood creatinine increased (Investigations) | 13 | 3
Neutrophil count decreased (Investigations) | 15 | 9
Weight decreased (Investigations) | 21 | 8
White blood cell count decreased (Investigations) | 16 | 13
Decreased appetite (Metabolism and nutrition disorders) | 56 | 46
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 16 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 10
Dizziness (Nervous system disorders) | 34 | 13
Dysgeusia (Nervous system disorders) | 45 | 17
Headache (Nervous system disorders) | 46 | 26
Neuropathy peripheral (Nervous system disorders) | 5 | 10
Paraesthesia (Nervous system disorders) | 13 | 7
Insomnia (Psychiatric disorders) | 19 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 29
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 35
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 7
Rash (Skin and subcutaneous tissue disorders) | 23 | 30
Neutropenia (Blood and lymphatic system disorders) | 41 | 18
Lacrimation increased (Eye disorders) | 1 | 9
Dysphagia (Gastrointestinal disorders) | 9 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 | 0
Pain (General disorders) | 10 | 9
Fall (Injury, poisoning and procedural complications) | 11 | 3
Electrocardiogram QT prolonged (Investigations) | 9 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 11 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 9 | 6
Visual perseveration (Nervous system disorders) | 12 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 | 8
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Bradycardia (Cardiac disorders) | 9 | 0

LIMITATIONS AND CAVEATS:
No analyses of ALK fusion variants or protein expression were done due to limited slide stability of unstained tissue sections required for immunohistochemistry and no nucleic acid based assay was available to identify specific ALK gene fusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.